
## The GlaxoSmithKline group of companies

203818

| Division | ŀ | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

Title : A Pilot Study to Evaluate Molecular Imaging Methods in Primary Sjögren's Syndrome : None

Effective Date : 08-JUN-2018

## **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 203818.
- This RAP will be provided to the study team members to convey the content of the final Statistical Analysis Complete (SAC) deliverable.

#### **Author's Name and Functional Area:**

| PPD | | 20 Apr 2019 |
|----------------|----------------------|-------------|
| Statistician ( | Clinical Statistics) | 20-Apr-2018 |

Copyright 2018 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# The GlaxoSmithKline group of companies

# **RAP Team Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| Principal Programmer (II Clinical Programming) | 31-MAY-2018 | PharmaTMF |
| Clinical Study Lead, Physician, RD II DPU | 25-MAY-2018 | PharmaTMF |
| Operations and Science Lead (II Clinical Pharmacology Science and Study Operations) | 31-MAY-2018 | PharmaTMF |
| Data Quality Leader (II Clinical Pharmacology<br>Science and Study Operations) | 25-MAY-2018 | PharmaTMF |
| (Imaging Lead, II TA) | 01-JUN-2018 | Email approval |
| (Molecular Imaging Consultant) | 07-JUN-2018 | Email approval |
| (Clinical Image Analysis) | 04-JUN-2018 | Email approval |
| Biologist, Research Manager in Transitional Sciences, DPU Lymphocyte Memo | 25-MAY-2018 | Email approval |

# **Clinical Statistics and Clinical Programming Line Approvals:**

| PPD | 00 HIN 2010 |
|--------------------------------|-------------|
| Director (Clinical Statistics) | 08-JUN-2018 |
| PPD | 07 HIN 2019 |
| Programming Manager | 07-JUN-2018 |

# **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | REPORTING | & ANALYSIS PLAN SYNOPSIS | 5 |
| 2. | <ul><li>2.1. Change</li><li>2.2. Study</li><li>2.3. Study</li></ul> | DF KEY PROTOCOL INFORMATIONges to the Protocol Defined Statistical Analysis Plan | 7<br>7 |
| 3. | <ul><li>3.1. Interin</li><li>3.2. Samp</li></ul> | NALYSES n Analyses le Size Re-estimation or Adjustment Analyses | 11<br>12 |
| 4. | | OPULATIONS | |
| 5. | | TIONS FOR DATA ANALYSES AND DATA HANDLING | 14 |
| 6. | | ULATION ANALYSESiew of Planned Analyses | |
| 7. | 7.1. Imagii<br>7.1.1.<br>7.1.2.<br>7.1.3. | 7.1.1.1. <sup>18</sup> F-FDG PET/CT | 16<br>17<br>17<br>18<br>18<br>19<br>19<br>20 |
| 8. | 8.1. Overv | ALYSESiew of Planned Adverse Events Analysesiew of Planned Clinical Laboratory Analyses | 21 |
| 9. | | 9.1.1.1. Comparison of pSS subjects with HV | 23<br>23<br>26 |
| 10. | REFERENCE | ES | 27 |


| 11. | APPE | NDICES | | 28 |
|---|---|---|---|---|
| | 11.1. | Appendix | x 1 : Time & Events | 29 |
| | 11.2. | Appendix | x 2: Data Display Standards & Handling Conventions | 31 |
| | | 11.2.1. | | |
| | | 11.2.2. | Baseline Definition & Derivations | 31 |
| | | | 11.2.2.1. Baseline Definitions | 31 |
| | | | 11.2.2.2. Derivations and Handling of Missing Baseline | |
| | | | Data | 31 |
| | | 11.2.3. | Reporting Process & Standards | 31 |
| | 11.3. | Appendix | x 3: Derived and Transformed Data | |
| | | 11.3.1. | General | 34 |
| | | 11.3.2. | Study Population | 34 |
| | | 11.3.3. | Imaging | 34 |
| | | 11.3.4. | Disease Activity Index | 35 |
| | | 11.3.5. | Histology | 41 |
| | | 11.3.6. | Laboratory Biomarkers of Disease Activity | 41 |
| | | 11.3.7. | Salivary Flow Rate | 42 |
| | | 11.3.8. | Lacrimal Function | 43 |
| | 11.4. | Appendix | x 4: Premature Withdrawals & Handling of Missing Data | 44 |
| | | 11.4.1. | | |
| | | 11.4.2. | Handling of Missing Data | 44 |
| | | | 11.4.2.1. Handling of Missing Dates | 44 |
| | | | 11.4.2.2. Handling of Partial Dates | 44 |
| | | | 11.4.2.3. Handling of Missing Data for Statistical | |
| | | | Analysis | 45 |
| | 11.5. | Appendix | x 5: Values of Potential Clinical Importance | 46 |
| | | 11.5.1. | Vital Signs | 46 |
| | | 11.5.2. | Laboratory Values | 46 |
| | 11.6. | | x 6: Multicentre Studies | |
| | 11.7. | | x 7: Examination of Covariates, Subgroups & Other Strata | |
| | 11.8. | | x 8: Multiple Comparisons & Multiplicity | 49 |
| | 11.9. | Appendix | x 9: Model Checking and Diagnostics for Statistical | |
| | | Analyses | S | 50 |
| | | 11.9.1. | Statistical Analysis Assumptions | 50 |
| | 11.10. | Appendix | x 10 – Abbreviations & Trade Marks | 51 |
| | | 11.10.1. | Abbreviations | 51 |
| | | 11.10.2. | Trademarks | 52 |
| | 11.11. | Appendix | x 11: List of Data Displays | 53 |
| | | | Data Display Numbering | |
| | | | Mock Example Shell Referencing | |
| | | | Deliverable [Priority] | |
| | | | Study Population Tables | |
| | | | Pharmacodynamic Tables | |
| | | 11.11.6. | Pharmacodynamic Figures | 59 |
| | | | Pharmacokinetic Tables | |
| | | | Pharmacokinetic Figures | |
| | | 11.11.9. | Safety Tables | 65 |
| | | | Biomarker Tables | |
| | | | .Biomarker Figures | |
| | | | LICH Listings | |
| | | | Non-ICH Listings | |
| | 11.12. | Appendix | x 12: Example Mock Shells for Data Displays | 83 |

# 1. REPORTING & ANALYSIS PLAN SYNOPSIS

| Overview | Key Elements of the RAP |
|---|---|
| Purpose | The purpose of this reporting and analysis plan (RAP) is to describe all planned analyses and outputs required for the final Clinical Study Report (CSR) of the study 203818. |
| Protocol | This RAP is based on the protocol amendment 1 [(Dated: 24/MAY2017) of study 203818 (GSK Document No.: 2015N227551_01] and eCRF Version 1. |
| Primary<br>Objective | To investigate the use of <sup>18</sup> F-FDG PET/CT in assessing increased glucose uptake as a biomarker of inflammation in pSS subjects. |
| | To investigate the use of <sup>11</sup> C- MET PET/CT in assessing salivary glandular function in pSS subjects and healthy volunteers. |
| | To investigate the use of multi-parametric MRI in assessing salivary gland inflammation, function and structure in pSS subjects and healthy volunteers. |
| Primary<br>Endpoint | Semi-quantitative parameters of uptake in selected body areas, including salivary glands for <sup>18</sup> F-FDG: |
| | - Standardised Uptake Value (SUV). |
| | - Tissue-to-reference (T/R) ratio. |
| | - Total inflammatory volume (TIV) where anatomically relevant. |
| | Semi-quantitative parameters of uptake in selected areas, including salivary glands for <sup>11</sup> C-MET: |
| | - SUV |
| | - T/R ratio |
| | - TIV where anatomically relevant. |
| | <ul> <li>Quantitative parameters of uptake derived from multi-parametric MRI in the<br/>salivary glands including: Exchange rate (K<sub>trans</sub>), Apparent Diffusion<br/>Coefficient (ADC), pure diffusion coefficient (D) and microvascular volume<br/>fraction (f) as data permits.</li> </ul> |
| Study<br>Design | This is an imaging study using PET/CT and multi parametric MRI to investigate the potential to characterise and quantify disease manifestation in pSS subjects, not involving therapeutic intervention. |
| | A minimum of 4 and up to 12 healthy volunteers will be enrolled in Group A (up to 8 subjects for <sup>11</sup> C-MET PET/CT imaging, up to 12 for MRI) and 8 to 12 pSS subjects will be enrolled in Group B. |
| | <ul> <li>Group A (healthy volunteers) will undergo an MRI of the salivary glands<br/>and <sup>11</sup>C-MET PET/CT (dynamic scan of the salivary glands followed by<br/>head to hip static scan).</li> </ul> |
| | Group B (pSS subjects) will undergo an MRI of the salivary glands, <sup>11</sup> C- |

| Overview | Key Elements of the RAP |
|---|---|
| | MET PET/CT (as for Group A) and <sup>18</sup> F-FDG PET/CT (head to hip). |
| Planned | <ul> <li>Interim analyses are detailed within Section 3.1 where applicable.</li> </ul> |
| Analyses | <ul> <li>All decisions regarding final analysis, as defined in this RAP document, will<br/>be made prior to Database Freeze of the study data.</li> </ul> |
| Analysis<br>Populations | The Screened Population (Comprises of subjects who sign the Informed Consent) will be used for the evaluation of Screen Failure subjects |
| | <ul> <li>The Safety Population (Comprised of all subjects who receive/undergo any<br/>Visit 1 procedure). will be used for the evaluation of Study Population and<br/>Safety.</li> </ul> |
| | The Pharmacokinetic (PK) Population (Comprised of subjects in the 'Safety' population for whom radio-pharmacokinetic sample was obtained and analysed) will be used for the evaluation of Pharmacokinetic Analysis. |
| Hypothesis | There are no formal hypotheses being tested in the study; instead an estimation and inference approach will be adopted to evaluate the objectives. |
| Primary<br>Analyses | Descriptive statistics and graphical displays, if appropriate, will be presented for all FDG PET/CT derived parameters across the regions of interest (ROI) for all pSS subjects and for all ¹¹C-MET PET/CT and MRI derived parameters across the ROI for all healthy volunteers and pSS subjects. |
| | <ul> <li>An exploratory comparison of pSS subjects vs healthy volunteers may be<br/>performed for each <sup>11</sup>C-MET PET/CT and MRI derived quantitative<br/>parameter as data permit, to estimate a difference (or ratio if log<br/>transformation is needed) with 95% confidence interval.</li> </ul> |
| Secondary<br>Analyses | Descriptive statistics and graphical displays, if appropriate, will also be presented for all derived parameters from dynamic PET imaging and PK analyses. |
| | If data permits, statistical analyses of <sup>11</sup> C-MET PET radio-PK modelling indices with <sup>11</sup> C-MET static imaging matrices will be conducted to assess correlation. |

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

There were no changes or deviations to the originally planned statistical analysis specified in the protocol [(Dated: 24/MAY/2017)]. However, the following objective has been added as this was not included in the protocol:

| Objectives | Endpoints |
|---|---|
| Exploratory Objectives | Exploratory Endpoints |
| To assess the safety and tolerability of study procedures, including <sup>18</sup> F-FDG PET/CT (pSS only), <sup>11</sup> C- MET PET/CT, multiparametric MRI and salivary gland biopsy (pSS only). | Safety and tolerability (Haematology, Clinical<br>Chemistry, Vital Signs, Adverse Events) |

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To investigate the use of <sup>18</sup> F-FDG PET/CT in assessing increased glucose uptake as a biomarker of inflammation in pSS subjects. | <ul> <li>Semi-quantitative parameters of uptake in selected body areas, including salivary glands for <sup>18</sup>F-FDG:</li> <li>Standardised Uptake Value (SUV)</li> <li>Tissue-to-reference ratio</li> <li>Total Inflammatory Volume (TIV) where anatomically relevant.</li> </ul> |
| To investigate the use of <sup>11</sup> C-MET PET/CT in assessing salivary glandular function in pSS subjects and healthy volunteers. | <ul> <li>Semi-quantitative parameters of uptake in selected areas, including salivary glands for <sup>11</sup>C-MET:</li> <li>Standardised Uptake Value (SUV)</li> <li>Tissue-to-reference ratio</li> <li>Total Inflammatory Volume (TIV) where anatomically relevant.</li> </ul> |
| To investigate the use of multi-<br>parametric MRI in assessing<br>salivary gland inflammation,<br>function and structure in pSS<br>subjects and healthy volunteers. | Quantitative parameters of uptake derived from multi-parametric MRI in the salivary glands including: Exchange rate (K <sub>trans</sub> ), Apparent Diffusion Coefficient (ADC), pure diffusion coefficient (D) and microvascular volume fraction (f) as data permits. |
| Secondary Objectives | Secondary Objectives |
| To characterize the pharmacokinetics of <sup>11</sup> C-MET PET tracer <i>in vivo</i> to allow static imaging parameters to be verified. | <ul> <li>Generation of quantitative outcome parameters<br/>(rate of <sup>11</sup>C-MET accumulation, as data permits)<br/>using a full quantitative analysis of dynamic PET<br/>scans.</li> <li>Comparison of static and dynamic imaging metrics</li> </ul> |

| Objectives | Endpoints |
|---|---|
| | in <sup>11</sup> C-MET. |
| Exploratory Objectives | Exploratory Objectives |
| To explore the use of novel multi-<br>parametric MRI in assessing<br>salivary gland inflammation,<br>function and structure in pSS<br>subjects and healthy volunteers. To explore the associations of the | Quantitative parameters of uptake derived from multi-parametric MRI in the salivary glands including, Initial Rate of Enhancement (IRE), maximal signal intensity enhancement (ME), lipid content, T1 relaxation and volume, as data permits. Association between 18E EDC DET/CT (necessity). |
| To explore the associations of the salivary gland imaging parameters with clinical and histological parameters of salivary glands. | <ul> <li>Association between <sup>18</sup>F-FDG PET/CT (pSS subjects only), <sup>11</sup>C-MET PET/CT and MRI parameters (healthy volunteers and pSS subjects) in the region of the salivary glands with each other and with clinical measures including: <ul> <li>Basal and stimulated salivary flow</li> <li>Histological scores from minor salivary gland biopsies including but not limited to lymphocyte count and focus score (pSS subjects)</li> <li>Laboratory biomarkers of disease activity (including metabolomic and/or proteomic profiles where applicable)</li> <li>European League Against Rheumatism (EULAR) Sjögren's Syndrome Disease Activity Index (ESSDAI) and EULAR Sjögren's Syndrome Patient Reported Index (ESSPRI), in particular subcomponents relevant to salivary gland function (pSS subjects).</li> </ul> </li> </ul> |
| To explore the extent of non-salivary gland (systemic) abnormalities detected on <sup>18</sup> F-FDG PET/CT and <sup>11</sup> CMET PET/CT, and the association of these abnormalities with clinical scores/relevant sub-scores and laboratory biomarkers in pSS subjects. | <ul> <li>Semi-quantitative parameters in selected areas systemically for <sup>18</sup>F-FDG and <sup>11</sup>C-MET (including but not limited to lymph nodes, thyroid, lacrimal glands, lungs and pancreas) and the associations of these parameters with: <ul> <li>Laboratory biomarkers of disease activity (including metabolomic and/or proteomic profiles where applicable)</li> <li>Lacrimal gland function as measured by Schirmer's test</li> <li>ESSDAI and ESSPRI and organ-specific subcomponents relating to the area imaged, where available.</li> </ul> </li> </ul> |
| To compare the metabolomic profiles of pSS subjects and healthy volunteers, to assess the intra-individual variability of the metabolome over time, and the ability of samples from different bodily sites to discriminate pSS | <ul> <li>Compare the metabolome/proteome of pSS subjects with healthy volunteers.</li> <li>Assess the variability in the metabolome and/or proteomic profile of individual subjects taken at 2 separate time points (Baseline and Visit 2).</li> <li>Compare the metabolome and/or proteomic profile from different body fluids/sites, and their utility in</li> </ul> |


| Objectives | Endpoints |
|---|---|
| subjects from healthy volunteers. | distinguishing pSS subjects from healthy volunteers. • Samples collected will be saliva, tears and plasma. |
| To assess the safety and tolerability of study procedures, including <sup>18</sup> F-FDG PET/CT (pSS only), <sup>11</sup> C- MET PET/CT, multiparametric MRI and salivary gland biopsy (pSS only). | Safety and tolerability (Haematology, Clinical<br>Chemistry, Vital Signs, Adverse Events) |

## 2.3. Study Design



| Overview of Study Design a | nd Key Features |
|---|---|
| | <ul> <li>Visit 2 should occur within 3 weeks after Visit 1. Visit 2 will involve measurement of basal and stimulated (chewing paraffin) salivary flow rate (including saliva collection), Schirmer's test (including tear collection), and blood samples for metabolomics/proteomics. In addition, a minor salivary gland biopsy will be performed on the pSS subjects (Group B).</li> <li>Visit 1 and Visit 2 may be split over more than one day.</li> </ul> |
| Contrast | <ul> <li><sup>18</sup>F-FDG (Group B only) radiotracer injected prior to PET/CT scanning.</li> <li><sup>11</sup>C-MET radiotracer injected prior to PET/CT scanning.</li> <li>Gadoterate meglumine (Dotarem®) contrast agent administered prior to MRI scanning</li> </ul> |
| Tracer Assignment | <ul> <li>All subjects will undergo MRI and <sup>11</sup>C-MET PET/CT at study visit 1.</li> <li>pSS subjects (Group B) will also undergo <sup>18</sup>F-FDG PET/CT at study visit 1.</li> </ul> |

# 2.4. Statistical Hypotheses

This study is designed to explore the use of <sup>18</sup>F-FDG PET/CT, <sup>11</sup>C-MET PET/CT, and multi-parametric MRI in pSS subjects and/or healthy volunteers. Due to the exploratory nature of this study, there are no formal hypotheses being tested, however exploratory comparisons may be conducted as outlined below:

For <sup>11</sup>C-MET PET/CT and multi-parametric MRI, pSS subjects will be compared to healthy volunteers using an estimation approach, providing point estimates of differences (or ratios as applicable) with 95% confidence intervals.

Descriptive summary tables and graphical plots will be used to summarise all the imaging parameters, if data permits.

## 3. PLANNED ANALYSES

## 3.1. Interim Analyses

No formal interim analysis will be performed. However, informal reviews of the imaging parameters will be performed to guide the decision to increase the sample size for one or more imaging modalities depending on the variability of the data, as described in the Interim Decision Document.

## 3.2. Sample Size Re-estimation or Adjustment

This is detailed in the Interim Decision Document.

## 3.3. Final Analyses

The final planned analyses will be performed after the completion of the following sequential steps:

- 1. All subjects have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release and database freeze has been declared by Data Management.

## 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Screened | Comprises of subjects who sign the<br>Informed Consent | Screen Failures |
| Safety | Comprised of all subjects who receives/undergoes any procedure on or after visit 1. | <ul> <li>Study Population</li> <li>Safety</li> <li>PET/CT Parameters</li> <li>Multiparametric-MRI Parameters</li> <li>Biomarkers</li> <li>Histological scores</li> <li>ESSDAI/ESSPRI</li> <li>Physician and patient global assessments, ocular and oral numerical rating scales</li> <li>Tear flow</li> <li>Salivary (basal and stimulated) flow</li> </ul> |
| Pharmacokinetic (PK) | Subjects in the 'Safety' population for whom<br>a radio-pharmacokinetic sample was<br>obtained and analysed. | <ul> <li>PET/CT radio-PK Concentrations</li> <li>Dynamic <sup>11</sup>C-MET PET/CT metrics</li> </ul> |

#### NOTES:

 Please refer to Appendix 11: List of Data Displayswhich details the population to be used for each display being generated.

#### 4.1. Protocol Deviations

• Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be listed.

- Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.
  - Data will be reviewed prior to freezing the database to ensure all important deviations and deviations which may lead to exclusion from the analysis are captured and categorised on the protocol deviations dataset.
  - o This dataset will be the basis for the listings of protocol deviations.
- A separate listing of all inclusion/exclusion criteria deviations will also be provided.
  This listing will be based on data as recorded on the inclusion/exclusion page of the
  eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

Table 1 provides an overview of appendices within the RAP for outlining general considerations for data analyses and data handling conventions.

Table 1 Overview of Appendices

| Section | Component |
|---|---|
| General ( | Considerations for Data Analyses & Data Handling Conventions |
| 11.1 | Appendix 1: Time & Events |
| 11.2 | Appendix 2: Data Display Standards & Handling Conventions |
| 11.3 | Appendix 3: Derived and Transformed Data |
| 11.4 | Appendix 4: Premature Withdrawals & Handling of Missing Data |
| 11.5 | Appendix 5: Values of Potential Clinical Importance |
| 11.6 | Appendix 6: Multicentre Studies |
| 11.7 | Appendix 7: Examination of Covariates, Subgroups & Other Strata |
| 11.8 | Appendix 8: Multiple Comparisons & Multiplicity |
| 11.9 | Appendix 9: Model Checking and Diagnostics for Statistical Analyses |
| Other RA | P Appendices |
| 11.10 | Appendix 10 – Abbreviations & Trade Marks |
| 11.11 | Appendix 11: List of Data Displays |
| 11.12 | Appendix 12: Example Mock Shells for Data Displays |

## 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Analyses

The study population analyses will be based on the Safety population. Screen failures will be listed based on the "Screened" population.

Table 2 provides an overview of the planned study population analyses, with full details of data displays being presented in Appendix 11: List of Data Displays

 Table 2
 Overview of Planned Study Population Analyses

| Endpoint / Parameter / Display Type | Data Display | s Generated |
|---|---|---|
| | Table | Listing |
| Subject Disposition | • | |
| Subject Disposition | Yes | |
| Reasons for Screen Failure | | Yes |
| Subjects by Centre | Yes | |
| Reasons for Study Withdrawal | | Yes |
| Protocol Deviations | • | |
| Important Protocol Deviations | | Yes |
| Subjects with Inclusion/Exclusion Criteria Deviations | | Yes [1] |
| Populations Analysed | | |
| Study Populations and Exclusions | Yes | |
| Subjects Excluded from Any Population | | Yes |
| Demographic and Baseline Characteristics | | |
| Demographic Characteristics | Yes | Yes |
| Race and Racial Combinations | Yes | Yes [2] |
| History of Tobacco Use | | Yes |
| Prior and Concomitant Medications | | |
| Current and Past Medical Conditions | | Yes |
| Concomitant Medications | Yes | Yes |
| Primary Sjogren's Syndrome History | | Yes |

#### NOTES:

- [1] Listing also includes analysis population exclusions.
- [2] Listing of race.

## 7. PRIMARY STATISTICAL ANALYSES

## 7.1. Imaging Analyses

## 7.1.1. Overview of Planned Imaging Analyses

The imaging analyses will be based on the Safety population, unless otherwise specified.

Table 3 provides an overview of the planned imaging analyses, with full details of data displays being presented in Appendix 11: List of Data Displays.

Table 3 Overview of Planned Imaging Analyses

| Endpoint / Parameter | Untransformed | | | | | | |
|---|---|---|---|---|---|---|---|
| | St | tats Analysi | S | Summary | | Individual | |
| | T | F | L | T | F | F | L |
| 18F-FDG PET/CT semi-quanti | tative pa | rameters | | | | | |
| SUV(mean/max/peak), T/R Ratio, TIV | | | | Yes <sup>1</sup> | Yes <sup>1</sup> | Yes <sup>1</sup> | Yes <sup>1</sup> |
| <sup>11</sup> C-MET PET/CT semi-quant | itative p | arameters | | | | | |
| SUV(mean/max/peak), T/R Ratio, TIV | Yes <sup>3</sup> | Yes <sup>3</sup> | | Yes <sup>2</sup> | | Yes <sup>2</sup> | Yes <sup>2</sup> |
| Multiparametric MRI quantitative parameters | | | | | | | |
| K <sub>trans</sub> <sup>4</sup> , ADC <sup>4</sup> , D <sup>4</sup> and f <sup>4</sup> | Yes <sup>3</sup> | Yes <sup>3</sup> | | Yes <sup>2</sup> | | Yes <sup>2</sup> | Yes <sup>2</sup> |

#### NOTES:

- T = Table, F = Figure, L = Listing
- SUV = Standard Uptake Value, T/R Ratio = Tissue-to-reference ratio, TIV = Total Inflammatory Volume (TIV), K<sub>trans</sub> = Exchange rate, ADC = Apparent Diffusion Coefficient, f = Microvascular volume fraction D = Pure Diffusion Coefficient
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- 1: By region of interest (ROI)
- 2: By region of interest (ROI) and group (Healthy Volunteers (HV) or primary Sjogren's Syndrome (pSS) patient).
- 3: If data permits. Stats analysis for SUV<sub>mean/max/peak</sub> for <sup>11</sup>C-MET PET/CT and K<sub>trans</sub>, D and f for MRI.
- 4: Median and IQR (Interguartile Range ) values for each parameter will be used.

#### 7.1.1.1. <sup>18</sup>F-FDG PET/CT

Descriptive statistics will be calculated and presented graphically and in tabular format for <sup>18</sup>F-FDG semi-quantitative derived parameters including SUV, Tissue-to-reference ratio and TIV (as data permits). All parameters will be listed by ROI (where ROI will be sorted by relevance to pSS subjects and ordered as Parotid gland, lacrimal, submandibular and lastly any other gland in alphabetical order). When applicable for a given ROI, the outputs will be separated by the side of the ROI having higher parameter values and lower parameter values. Aggregated measures (left-right combined) will use measures extracted over the combined ROI's, rather than left-right averages to not introduce a bias towards the smaller gland.

The data may be further explored using scatter plots to examine asymmetry in parameter values between left and right parotid glands.

Further details are given in Appendix 11: List of Data Displays.

#### 7.1.1.2. <sup>11</sup>C-MET PET/CT

Statistical analysis comparing the subject group (HV or pSS patient) will be conducted for  $^{11}$ C-MET PET/CT parameters (including but not limited to SUV<sub>mean</sub>, SUV<sub>max</sub> and SUV<sub>peak</sub>, as data permit), see Section 7.1.2 for detail.

Descriptive statistics will be calculated and presented graphically and in tabular format for <sup>11</sup>C-MET semi-quantitative derived parameters including SUV, Tissue-to-reference ratio and TIV and size of abnormality (as data permits). All parameters will be listed by group (HV or pSS patient) and ROI (where ROI will be sorted by relevance to pSS subjects and ordered as Parotid gland, lacrimal, submandibular and lastly any other gland in alphabetical order). When applicable for a given ROI, the analysis and summary outputs will be separated by the side of the ROI having higher parameter values and lower parameter values. Aggregated measures (left-right combined) will use measures extracted over the combined ROI's, rather than left-right averages to not introduce a bias towards the smaller gland.

The data may be further explored using scatter plots to examine asymmetry in parameter values between left and right parotid glands.

Further details are given in Appendix 11: List of Data Displays.

## 7.1.1.3. Multiparametric MRI

Statistical analysis comparing the subject group (HV or pSS patient) will be conducted for Multiparametric parameters (including but not limited to  $K_{trans}$ , D and f, as data permit), see Section 7.1.2 for detail. The median values of these parameters will be used for analysis.

Descriptive statistics will be calculated and presented graphically and in tabular format for multiparametric MRI quantitative derived parameters including but not limited to (median and IQR)  $K_{trans}$ , (median and IQR) ADC, (median and IQR) pure diffusion coefficient (D), and (median and IQR) microvascular fraction (f) as data permits. All parameters will be listed by group (HV or pSS patient) (and ROI, if data permits). When applicable for a given ROI, the analysis and summary outputs will be separated by the side of the ROI having higher parameter values and lower parameter values, as well as aggregated value. Aggregated measures (left-right combined) will use measures extracted over the combined ROI's, rather than left-right averages to not introduce a bias towards the smaller gland. As some of the MRI sequences may capture a reduced field-of-view of the salivary glands, the fraction of each gland that is analysed may be reported.

The data will be further explored using scatter plots and line plots to examine asymmetry in parameter values between left and right glands

Further details are given in Appendix 11: List of Data Displays.

## 7.1.1.4. Comparison of pSS subjects with HV

An exploratory comparison of pSS vs HV may be performed for <sup>11</sup>C-MET PET/CT and multiparametric MRI derived parameters as data permit, to estimate a difference (or ratio if log transformation is needed) with 95% confidence interval obtained from the analysis described in Section 7.1.2.

# 7.1.2. Planned Imaging Statistical Analyses

# **Primary Statistical Analyses**

## Endpoint(s)

- 11C-MET PET/CT derived parameters, including but not limited to SUV<sub>peak</sub>, SUV<sub>mean</sub>, SUV<sub>max</sub>
- Multiparametric MRI derived parameters, including but not limited to (median and IQR) K<sub>trans</sub>, (median and IQR) Pure diffusion coefficient (D), (median and IQR) microvascular volume fraction (f) and (median and IQR) ADC.

### **Model Specification**

- Parameters will be statistically analysed individually using an Analysis of Variance (ANOVA) model.
- Terms fitted in the ANOVA model will include:
   Fixed categorical: Subject group (HV or pSS patient)

#### **Model Checking & Diagnostics**

• Refer to Appendix 9: Model Checking and Diagnostics for Statistical Analyses: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

- Estimates of Difference (pSS-HV) (or Ratio (pSS/HV) if log<sub>e</sub> transformed) and 95% confidence interval for the derived parameters will be presented by ROI<sup>1</sup>.
- Plots of means (difference or ratio) and 95% confidence interval from the model will be generated for each ROI.
- P-values will not be presented as formal hypothesis is not being tested. The interpretation will be based on point estimates and its precision (95% CI).

#### NOTES:

• [1]: When applicable for a given ROI, the analysis will be separated by the side of the ROI having higher parameter values and lower parameter values, and aggregated over both sides.

## 7.1.3. Bayesian Analysis

In addition, a Bayesian approach to the exploratory comparison of pSS vs HV analysis of the <sup>11</sup>C-MET PET/CT and multi-parametric MRI parameters will be used. The objective of this analysis is to allow interpretable probability statements for the difference in two groups.

For the endpoints defined in Section 7.1.2, the uncertainty of the endpoint will be described with probability density function  $p(\mu)$ , say, where ' $\mu$ ' represents the parameter.  $P(\mu)$  represents our 'prior belief', since very little is known about the distribution of such parameters, normal function is assumed to be suitable for the data. This will have an unknown mean and known variance taken from the raw data (i.e  $x_i \sim N(\mu_i, \sigma_i^2)$ ) where j is

the pSS patient group or the HV group). A weakly-informative (vague) conjugate Normal prior density function with mean zero and a large variance will be adopted for the group mean  $(P(\mu)=N(0,100^2)$ .

The endpoint from the study data will be used to gather evidence, which will be characterised via its likelihood function (derived from the relevant sampling distribution,  $l(x|\mu)$ , say, where 'x' stands for 'data' or in our case the parameter values).

This will lead to a Normal posterior density function for the endpoints of interest. Should the data not support a Normal likelihood function, alternative parametric forms, such as a log-Normal density, will be investigated.

Bayes' theorem will be applied to derive the posterior density function  $p(\mu_j, x_j)$ . PROC MCMC will be used for the analysis in SAS. The number of burn-in iterations will be at least 10,000 and the number of MCMC iterations, excluding the burn-in iterations will be at least 5000.

The posterior distribution for each endpoint will be summarised by region and group, including mean, median, SD, interquartile range and 95% credible interval based on highest posterior density (HPD) interval.

Samples from the posterior distribution for the group mean  $p(\mu_i, x_i)$  for the pSS patients and for the HV subjects will be used to determine the posterior distribution for the ratio and difference of group means (pSS patients to the HV subjects). The posterior distribution for the ratio and difference of group means will be summarised by region and endpoint. Plots for the mean and 95% credible interval for the posterior distribution of the group mean and the difference of group means will be presented for each endpoint and region. Samples from the posterior distribution of the ratio of group means will be used to determine the probability that the ratio of the endpoints in pSS patients to HV subjects exceed 1 for each endpoint and region. This will be repeated for other values to allow us to plot a graph of probability of exceeding a certain value, for ratios of 1, 1.5 and 2. The ratio will be given such that group expected to have lower uptake will be used at the reference (denominator).

## 7.2. Pharmacokinetic Analyses

## 7.2.1. Overview of Planned Radio-Pharmacokinetic Analyses

The radio-PK analyses will be based on the PK population, unless otherwise specified. Influx rate constant (Ki) will be used as the imaging metric for <sup>11</sup>C-MET dynamic scan.

Table 4 provides an overview of the planned Radio-PK analyses, with further details of data displays being presented in Appendix 11: List of Data Displays.

Table 4 Overview of Planned Radio-Pharmacokinetic Analyses.

| Endpoint / Parameter/ | | Untransformed <sup>1</sup> | | | |
|---|---|---|---|---|---|
| Display Type | Stats A | nalysis | Summary | Individual | |
| | Τ | F | T | F | L |
| Radioactivity concentra | ations (whole | e blood and | plasma) | | |
| static <sup>18</sup> F-FDG PET/CT | | | | | Yes |
| <sup>11</sup> C-MET PET/CT | | | Yes | Yes <sup>2,3</sup> | Yes |
| Radiopharmacokinetic | parameters | (11C-MET) | | | |
| Influx rate constant (Ki) | Yes <sup>3</sup> | Yes <sup>3</sup> | Yes | | Yes |
| Administration Volume | | | | | |
| Tracer and contrast | | | | | Yes |
| Meal Ingested | Meal Ingested | | | | |
| Totality of Meal | | | | | Yes |
| ingested | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listings
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- [1]: Loge transform if necessary
- [2]: By subject group for <sup>11</sup>C-MET
- [3]: Correlation between radioPK parameter (Ki) vs <sup>11</sup>C-MET PET/CT SUV<sub>peak/mean/max</sub> by the side of the gland with most/least uptake in and ROI.

## 7.2.2. Radiopharmacokinetic Parameters

#### 7.2.2.1. Deriving Radiopharmacokinetic Parameters

Derivation of the influx rate constant (Ki) is described in the PET data acquisition and analysis protocol and the derived endpoint will be received from Imanova.

#### 7.2.2.2. Statistical Analysis of Radiopharmacokinetic Parameters

Tracer concentrations in whole blood and plasma will be summarized and listed by subject groups for static <sup>18</sup>F-FDG and <sup>11</sup>C-MET and Dynamic <sup>11</sup>C-MET. Individual, concentration-time curves will be plotted. The radio-pharmacokinetic parameter Influx Rate Constant (K<sub>i</sub>) for <sup>11</sup>C-MET PET/CT will be summarized and listed by subject groups.

<sup>11</sup>C-MET Influx rate constant (Ki) from dynamic <sup>11</sup>C-MET PET/CT scan will be graphically compared to <sup>11</sup>C-MET static scan SUV<sub>peak/mean/max</sub> or parameters derived by normalization with blood or other references, in the salivary gland region using a scatter plot by subject group. In addition to this, the correlation will be calculated and summarised between these parameters to compare static and dynamic imaging metrics.

## 8. SAFETY ANALYSES

# 8.1. Overview of Planned Adverse Events Analyses

The Safety analyses will be based on the Safety population, unless otherwise specified. Table 5 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 11: List of Data Displays.

Table 5 Overview of Planned Adverse Event Analyses

| Endpoint / Parameter/ Display Type | | lute <sup>1</sup> |
|---|---|---|
| | Summary | Individual |
| | Table | Listing |
| Adverse Events (AEs) | | |
| All AEs by SOC | Yes | Yes |
| Common AEs by Overall Frequency <sup>2</sup> | Yes | |
| Subjects & No. of Occurrences of Common Non-Serious AEs by SOC and PT <sup>2</sup> | Yes | |
| Subject Numbers for Individual AEs | | Yes |
| Relationship Between AE SOCs, PT & Verbatim Text | | Yes |
| Serious and Other Significant AEs | | |
| Reasons for Considering as a Serious AE | | Yes |
| AEs Leading to Withdrawal from Study by Overall Frequency | Yes | Yes |
| Subjects and Number of Occurrences of Serious and Fatal Serious AEs | Yes | |

#### NOTES:

- SOC = System Organ Class, PT = Preferred Term.
- Summary = Represents TF related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- [1]: All outputs by subject group (HV and pSS)
- [2]: Common defined by ≥ 2 subjects

# 8.2. Overview of Planned Clinical Laboratory Analyses

The Clinical Laboratory analyses will be based on the "Safety" population, unless otherwise specified.

Table 6 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 11: List of Data Displays.

Table 6 Overview of Planned Clinical Laboratory Analyses

| Endpoint / Parameter/ Display Type | Absolute |
|------------------------------------|------------|
| | Individual |
| | Listing |
| Chemistry | |
| Chemistry | Yes |
| Hematology | Yes |
| Urinalysis | Yes |


203818

| Endpoint / Parameter/ Display Type | Absolute |
|---|---|
| | Individual |
| | Listing |
| Other Screening Tests | Yes |
| Vital Signs | |
| Vital Signs for Subjects with Values of Potential Clinical Importance (PCI) | Yes |

# NOTES:,

- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

## 9. OTHER STATISTICAL ANALYSES

# 9.1. Exploratory Analyses

# 9.1.1. Overview of Exploratory Analyses

The exploratory analyses will be based on the Safety population, unless otherwise specified.

Table 7 provides an overview of the planned exploratory analyses, with full details of data displays being presented in Appendix 11: List of Data Displays.

Table 7 Overview of Planned Exploratory Analyses

| Endpoint | Untransformed | | | | |
|---|---|---|---|---|---|
| | Absolute | | | | |
| | Sumi | | Individual | | Stats Analysis |
| | Т | F | F | L | T |
| Salivary gland | T | Т | Т | | 1 |
| Basal and Stimulated salivary flow | Yes | | Yes | Yes | Yes <sup>1</sup> |
| Histological scores <sup>2</sup> | Yes | | Yes | Yes | Yes <sup>1</sup> |
| Lacrimal Gland | | | | | |
| Schirmer's test | Yes | | Yes | Yes | Yes <sup>1</sup> |
| Disease index <sup>2</sup> | | | | | |
| Disease activity measures <sup>3</sup> | Yes | | | Yes | |
| ESSDAI and ESSPRI | | | Yes | | Yes <sup>1</sup> |
| ESSDAI component scores | Yes | | | Yes | |
| ESSPRI component scores | | | | Yes | |
| Multiparametric MRI quantitative param | neters <sup>5</sup> | | | | |
| (median and IQR) IRE, (median and | | | | | |
| IQR) ME, (mean) Lipid Content, | | | | | |
| (median and IQR) T1 relaxation, | Yes <sup>6</sup> | Yes <sup>6</sup> | | Yes <sup>6</sup> | Yes <sup>1, 7</sup> |
| (median and IQR) D* and (mean) gland | | | | | |
| volume | | | | | |
| Multiparametric MRI Questionnaire | | | | | |
| Dental History | | | | Yes | |
| Sjogren's specific biomarkers <sup>2</sup> | | | | | |
| Laboratory biomarkers of disease activity <sup>4</sup> | Yes | | Yes | Yes | Yes <sup>1</sup> |

#### NOTES:

- T = Table, F = Figure, L = Listing, IQR = Interquartile Range, D\* = Psuedo Diffusion
- Summary = Represents TFL related to any summaries (descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- 1: Summary table for correlation.
- 2: pSS subjects only more detail below
- 3: These include ESSDAI, ESSPRI, Patient Global Assessment, Physician Global Assessment, Oral dryness

numerical rating, ocular dryness numerical rating

- 4: This may include metabolomic and proteomic profiles if applicable and also include data from healthy subjects.
   See Section 11.3.6 for more details.
- 5: If data permits.
- 6: By region of interest (ROI) and group (HV or pSS patient).
- 7: Summary table of comparison between HV and pSS group.

Descriptive statistics (Mean, Median, Standard Deviation, Minimum, Maximum) of absolute values of basal, stimulated salivary flow rate and score from Schirmer's test will be provided. The absolute values will be listed by subject groups.

The histological scores (see Section 11.3.5) and the various disease indices (see Section 11.3.4) – ESSDAI, ESSPRI, Patient and Physician global assessment of disease activity, oral and ocular dryness scales will be descriptively summarized and listed for pSS group only.

Descriptive statistics will be calculated for the exploratory multiparametric MRI quantitative derived parameters listed in Table 7 (as data permits) and presented in tables. All parameters will be listed by group (and ROI, as data permits). Mean (± SE bars) will be plotted for each parameter by ROI (if appropriate with panel for each side).

Correlation between  $^{18}$ F-FDG PET/CT (pSS subjects only),  $^{11}$ C-MET PET/CT and MRI parameters (HV and pSS subjects) in the region of the salivary glands (parotid gland) will be explored using scatter plots. Plots will be in panel for each side (most vs least uptake) of the region scanned. The parameters will include,  $SUV_{peak}$  for PET/CT and  $K_{trans}$ , D and f for multiparametric MRI.

Furthermore, correlation between the imaging parameters mentioned above and

- histological scores (mean and maximum lymphoid organisation score and volume fraction) from the minor salivary gland biopsy
- Salivary flow rate mean (from baseline and visit 2) stimulated and basal salivary flow rate, and mean difference (stimulated basal)
- Measures of Disease Activity ESSDAI and ESSPRI scores
- Lab biomarkers of disease activity C3 and C4 levels
- Schirmer's test length of paper wetted by eyes (panel for each side; least and most) and time to completely wet the strip (panel for each side; least and most).

may be explored using scatter plots (panel for each side) and statistical analysis summarised in tables. In addition,  $SUV_{peak}$  from the  $^{11}C$ -MET PET/CT will be correlated with the ratio of IgG/IgA using scatter plots and summary tables of the correlation. See below for summary of correlations:

| Method | | 11C-MET PET/CT | 18F-FDG PET/CT | Multiparametric MRI |
|---|---|---|---|---|
| | Parameter(s)/Endpoint | SUVpeak | SUVpeak | (median) Ktrans, (median) D,<br>(median) ADC, (median) f,<br>(median) IRE, (median) ME,<br>(mean) Lipid Content, (median)<br>D* (pseudo diffusion), (mean)<br>gland volume |
| 11C-MET PET/CT | SUVpeak | | Yes | |
| 18F-FDG PET/CT | SUVpeak | Yes | | |
| Multiparametric<br>MRI | (mean) lipid content | Yes | Yes | Yes <sup>1</sup> |
| Histological scores | Max lymphocyte focus score | Yes | Yes | Yes |
| | Mean lymphocyte focus score | | | |
| | Max Lymphoid organisation grading | | | |
| | Mean Lymphoid organisation grading | | | |
| Salivary flow rate | Mean stimulated | Yes | Yes | Yes |
| | Mean basal | | | |
| | Mean difference | | | |
| Disease Activity | ESSDAI | Yes | Yes | Yes |
| | ESSPRI | | | |
| Lab biomarkers of | C3 | Yes | Yes | Yes |
| disease activity | C4 | | | |
| | IgG/IgA | Yes | Yes | Yes |
| Schirmer's test | Length wet per minute | Yes | Yes | |

<sup>[1]:</sup> Correlation of lipid content with (median) Ktrans, IRE, ME, D, f, ADC.

If metabolomic and/or proteomic data is available in the study, these may be reported as a separate reporting effort in addition to the final SAC reporting effort. This will not contribute to the CPSR.

## 9.1.1.1. Comparison of pSS subjects with HV

An exploratory comparison of pSS vs HV may be performed for multiparametric MRI derived exploratory parameters as data permit, to estimate a difference (or ratio if log transformation is needed) with 95% confidence interval obtained from the analysis described in Section 9.1.2.

## 9.1.2. Planned Imaging Statistical Analyses

# **Primary Statistical Analyses**

#### Endpoint(s)

 Multiparametric MRI derived parameters; (median and IQR) IRE, (median and IQR) ME, (mean) Lipid Content, (median and IQR) T1 relaxation, (median and IQR) D\* (pseudo diffusion) and (mean) gland volume

#### **Model Specification**

- Parameters will be statistically analysed using an Analysis of Variance (ANOVA) model.
- Terms fitted in the ANOVA model will include:
   Fixed categorical: Subject group (HV or pSS patient)

## **Model Checking & Diagnostics**

 Refer to Appendix 9: Model Checking and Diagnostics for Statistical Analyses: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

- Estimates of Difference (pSS-HV) (or Ratio (pSS/HV) if log<sub>e</sub> transformed) and 95% confidence interval for the derived parameters will be presented by ROI¹.
- Plots of means (difference or ratio) and 95% confidence interval from the model will be generated for each ROI.
- P-values will not be presented as formal hypothesis is not being tested. The interpretation will be based on point estimates and its precision (95% CI).

**NOTES:** [1]: When applicable for a given ROI, the analysis will be separated by the side of the ROI having higher parameter values and lower parameter values, and aggregated over both sides.

# 10. REFERENCES

Cho, H., Yoo, J., Yun, C., Kang, E., Lee, H., Hyon, J., Song, Y. and Lee, Y. (2013). The EULAR Sjogren's syndrome patient reported index as an independent determinant of health-related quality of life in primary Sjogren's syndrome patients: in comparison with non-Sjogren's syndrome patients. *Rheumatology*, 52(12), pp.2208-2217

GlaxoSmithKline Document Number 2015N227551\_01 Study ID 203818: A Pilot Study to Evaluate Molecular Imaging Methods in Primary Sjögren's Syndrome. 24-MAY-2018

#### Interim Decision Document

https://biodocumentum.bio.corpnet1.com/webtoppr/drl/objectId/090f45f68622127b (00\_No Asset-203818 Statistical Analysis Plan (Interim Decision Document) Version 001 (14-Sep-2017))

# 11. APPENDICES

| Section | Appendix |
|---|---|
| General Considerations for Data Analyses & Data Handling Conventions | |
| Section 11.1 | Appendix 1: Time & Events |
| Section 11.2 | Appendix 2: Data Display Standards & Handling Conventions |
| | Study Treatment & Sub-group Display Descriptors |
| | Baseline Definitions & Derivations |
| | Reporting Process & Standards |
| Section 11.3 | Appendix 3: Derived and Transformed Data |
| | General, Study Population & Safety |
| | Efficacy |
| | Pharmacokinetic |
| | Pharmacodynamic and or Biomarkers |
| Section 11.4 | Appendix 4: Premature Withdrawals & Handling of Missing Data |
| | Premature Withdrawals |
| | Handling of Missing Data |
| Section 11.5 | Appendix 5: Values of Potential Clinical Importance |
| Section 11.6 | Appendix 6: Multicentre Studies |
| Section 11.7 | Appendix 7: Examination of Covariates, Subgroups & Other Strata |
| Section 11.8 | Appendix 8: Multiple Comparisons & Multiplicity |
| Section 11.9 | Appendix 9: Model Checking and Diagnostics for Statistical Analyses |
| Other RAP App | endices |
| Section 11.10 | Appendix 10 – Abbreviations & Trade Marks |
| Section 11.11 | Appendix 11: List of Data Displays |
| Section 11.12 | Appendix 12: Example Mock Shells for Data Displays |

# 11.1. Appendix 1 : Time & Events

## Time and Events Table - Screening and Baseline Assessments

| Procedure | Screening/Baseline<br>Visit | Baseline 2<br>(FRP only) |
|---|---|---|
| | | Within 3-8 days prior to Visit 1 |
| Informed consent | X | |
| Inclusion and exclusion criteria | X | |
| Demography | X | |
| Medical history including past and current medical conditions | X | |
| Full physical exam (including height and weight) | X | |
| MRI safety questionnaire | X | |
| Vital signs | X | |
| Concomitant medication review | χ | |
| ESSDAI | <b>X</b> <sup>1</sup> | |
| ESSPRI | <b>X</b> <sup>1</sup> | |
| Oral dryness numerical rating | <b>X</b> <sup>1</sup> | |
| Ocular dryness numerical rating | <b>X</b> <sup>1</sup> | |
| Patient global assessment | <b>X</b> 1 | |
| Physician's global assessment | <b>X</b> 1 | |
| Basal salivary flow | Χ | |
| Stimulated salivary flow (including saliva collection) | X | |
| Schirmer's test (including tear collection) | X | |
| Plasma metabolomics/proteomics | X | |
| Haematology/clinical chemistry [ | X | |
| Blood biomarkers for ESSDAI | <b>X</b> 1 | |
| Autoantibody screen (anti-Sjögren's-syndrome- | | |
| related antigen A [Anti-SSa], anti Sjögren's | <b>X</b> <sup>1</sup> | |
| syndrome type B [SSb]) | | |
| FSH/oestradiol (post-menopausal women only) | χ | |
| Serum pregnancy test (FRP) | <b>X</b> <sup>2</sup> | |
| Urine pregnancy test( FRP) | | X <sup>2</sup> |
| Urinalysis | X3 | animar EDD – fermales of |

AE = adverse event; FSH = follicle stimulating hormone; MRI = magnetic resonance imaging; FRP = females of reproductive potential; .ESSDAI = European League Against Rheumatism (EULAR) Sjögren's Syndrome Disease Activity Index; ESSPRI = EULAR Sjögren's Syndrome Patient Reported Index

- 1. pSS subjects only
- 2. Females of reproductive potential only.
- 3. Urine to be sent for urine protein:creatinine ratio if ≥trace proteinuria by dipstick.

#### **Time and Events Table - Study Assessments**

| Procedure | Visit 1 | Visit 2 | Follow up |
|---|---|---|---|
| | Within 6 weeks after baseline | Within 3 weeks<br>after Visit 1 | Within 2 weeks after Visit 2 |
| MRI safety questionnaire <sup>5</sup> | Х | | |
| Vital signs | Х | Х | |
| Concomitant medication review | Х | Х | |
| Basal salivary flow | | Х | |
| Stimulated salivary flow (including saliva | | Х | |
| collection) | | | |
| Schirmer's test (including tear collection) | | Х | |
| Plasma metabolomics/proteomics | | Х | |
| Urine pregnancy test (FRP) | <b>X</b> 1 | <b>X</b> 1 | |
| Multi-parametric MRI scan (including | Х | | |
| contrast) | | | |
| Meal prior to <sup>11</sup> C-MET PET/CT | Х | | |
| Intravenous injection of <sup>11</sup> C-MET PET tracer | Х | | |
| <sup>11</sup> C-MET PET/CT scan (dynamic and static) | Х | | |
| Radio-PK (11C-MET) sampling (dynamic scan) | X <sup>2</sup> | | |
| Measure concentration of <sup>11</sup> C-MET tracer in | <b>X</b> 3 | | |
| blood | | | |
| Blood glucose (bedside glucometer) | Χ4 | | |
| Injection of <sup>18</sup> F-FDG tracer | Χ4 | | |
| <sup>18</sup> F-FDG PET/CT scan | Χ4 | | |
| Measure concentration of <sup>18</sup> F-FDG in blood | X3,4 | | |
| Salivary gland biopsy | | <b>X</b> 4 | |
| AE review | | Χ | |

AE = adverse event; CT = computed Tomography; FDG = flurodeoxyglucose; FRP = females of reproductive potential; FSH = follicle stimulating hormone; MET = methionine; MRI = magnetic resonance imaging; PET = positron emission tomography; PK = pharmacokinetics;.

- 1. Females of reproductive potential only
- 2. Radio-PK sampling (5mL per sample) to be taken at 1, 2, 5, 10, 15, 20, 30 and 40 minutes after injection of <sup>11</sup>C-MET PET tracer (number and sampling times are subject to change dependent on emerging data, but no more than 100 mL overall will be taken).
- 3. To be taken within 5 minutes after the static PET/CT scan (exact time to be recorded).
- 4. pSS subjects only. If it is not possible to schedule the minor salivary gland biopsy within the 3 week window after Visit 1, this procedure may be performed up to 6 weeks after Visit 1, subject to prior agreement of the medical monitor.
- 5. The MRI safety questionnaire will not be databased

# 11.2. Appendix 2: Data Display Standards & Handling Conventions

#### 11.2.1. Study Treatment Display Descriptors

No study treatment is administered in this study. Subject group displays will be described as follows:

| | Subject Group | Descriptions | |
|---|---|---|---|
| | Dataset Display Data Displays for Reporting | | ng |
| Code | Description | Description | Order [1] |
| Н | Healthy Volunteer | Healthy Volunteer | 1 |
| Р | pSS Patient | pSS Patient | 2 |

#### NOTES:

#### 11.2.2. Baseline Definition & Derivations

#### 11.2.2.1. Baseline Definitions

For all endpoints, baseline will be taken as the value at the screening/baseline except for urine pregnancy test which is taken at baseline 2 (within 4-7 days prior to Visit 1).

#### 11.2.2.2. Derivations and Handling of Missing Baseline Data

No change from baseline calculations are to be conducted. However, if required then the following derivation is to be used:

| | Reporting Details |
|----------------------|----------------------------------------------|
| Change from Baseline | = Post-Baseline Visit Value – Baseline Value |

#### NOTES:

- Unless otherwise specified, the baseline definitions specified in Section 11.2.2.1 Baseline Definitions will be used for derivations for endpoints / parameters and indicated on summaries and listings.
- Unless otherwise stated, if baseline data is missing no derivation will be performed and will be set to missing.
- The baseline definition will be footnoted on all change from baseline displays.

#### 11.2.3. Reporting Process & Standards

| Reporting Proces | s |
|---|---|
| Software | |
| The currently : | supported versions of SAS software will be used. |
| Reporting Area | |
| HARP Server | : UK1SALX00175 |
| HARP Area : /ARPROD/NOCOMPOUND/MID203818/FINAL | |

<sup>1.</sup> Order represents subject groups being presented in TFL, as appropriate.

| _ | | 4. | | _ | | |
|-----|----|---------|---|----|--------------|-----|
| Pο | nn | rtin | ~ | Ur | $\sim$ | 200 |
| 1/6 | ·u | /I LIII | u | | $\mathbf{v}$ | .55 |

QC Spreadsheet : /ARWORK/NOCOMPOUND/MID203818/FINAL/DOCUMENTS

#### **Analysis Datasets**

 Analysis datasets will be created according to Integrated Data Standards Library (IDSL) GSK A&R dataset standards.

#### **Generation of RTF Files**

RTF files will be generated for the final analysis tables and listings only.

## **Reporting Standards**

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated:
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- All data will be reported according to the actual treatment the subject received unless otherwise stated.
- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### Planned and Actual Time

- Reporting for tables, figures and formal statistical analyses:
  - For Imaging related outputs, the planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, where the output is radio-pharmacokinetic related. For any other outputs the planned time relative to visit 1.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - For Imaging related outputs, planned and actual time relative to study contrast administration will be shown in listings (Refer to IDSL Statistical Principle 5.05.1). For any other outputs, planned and actual time relative to Visit 1 will be shown in listings.
  - Unscheduled or unplanned readings will be presented within the subject's listings.
  - Visits outside the protocol defined time-windows (i.e. recorded as protocol deviations) will be included in listings but omitted from figures, summaries and statistical analyses.

#### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables.
- Unscheduled visits will not be included in figures.
- All unscheduled visits will be included in listings.


| Reporting Standards | |
|---|---|
| Descriptive Summary Statistics | |
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| <b>Graphical Displays</b> | Graphical Displays |
| Refer to IDSL St | atistical Principals 7.01 to 7.13. |

# 11.3. Appendix 3: Derived and Transformed Data

#### 11.3.1. **General**

#### **Multiple Measurements at One Time Point**

 Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.

#### **Study Day**

- Calculated as the number of days from Visit 1 date:
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < Visit 1 Date → Study Day = Ref Date Visit 1 Date
  - Ref Data ≥ Visit 1 Date → Study Day = Ref Date (Visit 1 Date) + 1

## 11.3.2. Study Population

#### **Demographics**

#### Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - Any subject with a missing date and month will have this imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.
- The reference day for age calculation will be screening visit.

## **Body Mass Index (BMI)**

Calculated as Weight (kg) / [Height (m)<sup>2</sup>]

## 11.3.3. Imaging

## **Imaging Parameters**

All imaging parameters datasets will contain ROI which will include the side of the ROI where applicable. A variable will be derived for the side with the higher (named 'High') and lower (named 'Low') parameter value. When ROI does not have a side or in the case where the sides have equal parameter values the variable will be 'NA'. The variable can be called 'Side', to aid with the reporting of the study. For MRI parameters, the aggregated score will be included for listing and summary tables and plots. No derivations will be conducted by GSK.

## 11.3.4. Disease Activity Index

#### **Disease Activity Index**

#### **ESSDAI**

The European League Against Rheumatism (EULAR) Sjögren's syndrome disease activity index (ESSDAI) is a systemic disease activity index that was designed to measure disease activity in patients with primary SS. The ESSDAI is a disease activity index that was generated in 2009, by consensus of a large group of worldwide experts from European and North American countries. The ESSDAI is a systemic diease activity index and includes 12 domains (i.e., organ systems; cutaneous, respiratory, renal, articular, muscular, peripheral nervous system (PNS), central nervous system (CNS), haematological, glandular, constitutional, lymphadenopathic, biological). Each domain is divided in three to four levels depending on their degree activity. The final score, the sum of all domain scores (given below), falls between 0 and theoretically 123, with 0 being no disease activity and 123 being most severe disease activity.

| Domain | Activity level | Description |
|---|---|---|
| Constitutional - Exclusion of fever | No=0 | Absence of the following symptoms |
| of infectious origin<br>and voluntary<br>weight loss | Low=3 | Mild or intermittent fever (37.5°–38.5°C)/night sweats and/or involuntary weight loss of 5–10% of body weight |
| | Moderate=6 | Severe fever (>38.5°C) / night sweats and/or involuntary weight loss of >10% of body weight |
| Lymphadenopathy - Exclusion of | No=0 | Absence of the following features |
| infection | Low=4 | Lymphadenopathy ≥1 cm in any nodal region or ≥2 cm in inguinal region |
| | Moderate=8 | Lymphadenopathy ≥2 cm in any nodal region or ≥3 cm in inguinal region, and/or splenomegaly (clinically palpable or assessed by imaging) |
| | High=12 | Current malignant B-cell proliferative disorder* |
| Glandular -<br>Exclusion of stone | No=0 | Absence of glandular swelling |
| or infection | Low=2 | Small glandular swelling with enlarged parotid (≤3 cm), or limited submandibular or lachrymal swelling |
| | Moderate=4 | Major glandular swelling with enlarged parotid (>3 cm), or important submandibular or lachrymal swelling |

| Articular - | No=0 | Absence of currently active articular |
|---|---|---|
| Exclusion of osteoarthritis | 110-0 | involvement |
| | Low=2 | Arthralgias in hands, wrists, ankles and feet accompanied by morning stiffness (>30 min) |
| | Moderate=4 | 1–5 (of 28 total count) synovitis |
| | High=6 | ≥6 (of 28 total count) synovitis |
| Cutaneous - Rate as 'No activity' stable long-lasting | No=0 | Absence of currently active cutaneous involvement |
| features related to damage | Low=3 | Erythema multiforma |
| uamage | Moderate=6 | Limited cutaneous vasculitis, including urticarial vasculitis, or purpura limited to feet and ankle, or subacute cutaneous lupus |
| | High=9 | Diffuse cutaneous vasculitis, including urticarial vasculitis, or diffuse purpura, or ulcers related to vasculitis |
| Pulmonary - Rate as 'No activity' stable long-lasting features related to damage, or respiratory involvement not related to the disease (tobacco use, etc.) | No=0 | Absence of currently active pulmonary involvement |
| | Low=5 | Persistent cough or bronchial involvement with no radiographic abnormalities on radiography Or radiological or HRCT evidence of interstitial lung disease with: No breathlessness and normal lung function test. |
| | Moderate=10 | Moderately active pulmonary involvement, such as interstitial lung disease shown by HRCT with shortness of breath on exercise (NHYA II) or abnormal lung function tests restricted to: $70\%$ >DL <sub>CO</sub> $\geq$ 40% or $80\%$ >FVC $\geq$ 60% |
| | High=15 | Highly active pulmonary involvement, such as interstitial lung disease shown by HRCT with shortness of breath at rest (NHYA III, IV) or with abnormal lung function tests: $DL_{CO} < 40\%$ or $FVC < 60\%$ |
| isease Activity Index | | |
|---|---|---|
| Renal - Rate as 'No activity' stable long-lasting features related to damage, and renal involvement not related to the disease. If biopsy has been performed, please rate activity based on histological features first | No=0 | Absence of currently active renal involvement with proteinuria <0.5 g/day, no haematuria, no leucocyturia, no acidosis, or long-lasting stable proteinuria due to damage |
| | Low=5 | Evidence of mild active renal involvement, limited to tubular acidosis without renal failure or glomerular involvement with proteinuria (between 0.5 and 1 g/day) and without haematuria or renal failure (GFR ≥60 mL/min) |
| | Moderate=10 | Moderately active renal involvement, such as tubular acidosis with renal failure (GFR <60 mL/min) or glomerular involvement with proteinuria between 1 and 1.5 g/day and without haematuria or renal failure (GFR ≥60 mL/min) or histological evidence of extra-membranous glomerulonephritis or important interstitial lymphoid infiltrate |
| | High=15 | Highly active renal involvement, such as glomerular involvement with proteinuria >1.5 g/day or haematuria or renal failure (GFR <60 mL/min), or histological evidence of proliferative glomerulonephritis or cryoglobulinemia related renal involvement |
| Muscular - Exclusion of weakness due to corticosteroids | No=0 | Absence of currently active muscular involvement |
| | Low=6 | Mild active myositis shown by abnormal EMG or biopsy with no weakness and creatine kinase (N <ck\le 2n)<="" td=""></ck\le> |
| | Moderate=12 | Moderately active myositis proven by abnormal EMG or biopsy with weakness (maximal deficit of 4/5), or elevated creatine kinase (2N < CK ≤ 4N), |
| | High=18 | Highly active myositis shown by abnormal EMG or biopsy with weakness (deficit ≤3/5) or elevated creatine kinase (>4N) |

| Disease Activity Index | | |
|---|---|---|
| PNS - Rate as 'No activity' stable long-lasting | No=0 | Absence of currently active PNS involvement |
| features related to damage or PNS involvement not related to the disease | Low=5 | Mild active peripheral nervous system involvement, such as pure sensory axonal polyneuropathy shown by NCS or trigeminal (V) neuralgia |
| | Moderate=10 | Moderately active peripheral nervous system involvement shown by NCS, such as axonal sensory-motor neuropathy with maximal motor deficit of 4/5, pure sensory neuropathy with presence of cryoglobulinemic vasculitis, ganglionopathy with symptoms restricted to mild/moderate ataxia, inflammatory demyelinating polyneuropathy (CIDP) with mild functional impairment (maximal motor deficit of 4/5or mild ataxia), |
| | | origin (except trigeminal (V) neuralgia) |
| | High=15 | Highly active PNS involvement shown by NCS, such as axonal sensory-motor neuropathy with motor deficit ≤3/5, peripheral nerve involvement due to vasculitis (mononeuritis multiplex, etc), severe ataxia due to ganglionopathy, inflammatory demyelinating polyneuropathy (CIDP) with severe functional impairment: motor deficit ≤3/5 or severe ataxia |
| CNS - Rate as 'No activity' stable long-lasting | No=0 | Absence of currently active CNS involvement |
| features related to<br>damage or CNS<br>involvement not<br>related to the<br>disease | Moderate=10 | Moderately active CNS features, such as cranial nerve involvement of central origin, optic neuritis or multiple sclerosis-like syndrome with symptoms restricted to pure sensory impairment or proven cognitive impairment |

| Disease Activity Index | | |
|---|---|---|
| · | High=15 | Highly active CNS features, such as cerebral vasculitis with cerebrovascular accident or transient ischaemic attack, seizures, transverse myelitis, lymphocytic meningitis, multiple sclerosis-like syndrome with motor deficit. |
| Haematological -<br>For anaemia, | No=0 | Absence of autoimmune cytopenia |
| neutropenia, and<br>thrombopenia, only<br>autoimmune<br>cytopenia must be<br>considered<br>Exclusion of<br>vitamin or iron<br>deficiency, drug-<br>induced cytopenia | Low=2 | Cytopenia of autoimmune origin with neutropenia (1000 <neutrophils<1500 (100="" (10<hae-ahaemoglobin<12="" (500<lymphocytes<1000="" 000="" 000<platelets<150="" anaemia="" and="" dl),="" g="" lymphopenia="" mm³)="" mm³),="" mm³)<="" or="" td="" thrombocytopenia=""></neutrophils<1500> |
| | Moderate=4 | Cytopenia of autoimmune origin with neutropenia (500\le neutrophils\le 1000/mm³), and/or anaemia (8\le haemoglobin\le 10 g/dL), and/or thrombocytopenia (50 000\le platelets\le 100 000/mm³) Or lymphopenia (\le 500/mm3) |
| | High=6 | Cytopenia of autoimmune origin with neutropenia (neutrophils <500/mm³), and/or or anaemia (haemoglobin <8 g/dL) and/or thrombocytopenia (platelets <50 000/mm³) |
| Biological | No=0 | Absence of any of the following biological features |
| | Low=1 | Clonal component and/or<br>hypocomplementemia (low C4 or C3 or<br>CH50) and/or hypergammaglobulinemia or<br>high IgG level between 16 and 20 g/L |
| | Moderate=2 | Presence of cryoglobulinemia and/or hypergammaglobulinemia or high IgG level >20 g/L, and/or recent onset hypogammaglobulinemia or recent decrease of IgG level (<5 g/L) |

| Disease Activity Index |
|---|
| ESSPRI |
| The EULAR Sjögren's syndrome patient reported index (ESSPRI) was developed as a simple index for measuring pSS patient's symptoms. The ESSPRI is calculated by averaging the scales for pain, fatigue and dryness (Cho et al., 2013). The final ESSPRI score is therefore continuous and ranges from 0 to 10 with 10 being maximal pSS symptoms. |
| 1) How severe has your dryness been during the last 2 weeks? |
| No Maximal imaginable dryness 0 1 2 3 4 5 6 7 8 9 10 Maximal imaginable dryness |
| 2) How severe has your fatigue been during the last 2 weeks? |
| No fatigue 0 1 2 3 4 5 6 7 8 9 10 Maximal imaginable fatigue |
| 3) How severe has your pain (joint or muscular pains in your arms or legs)<br>been during the last 2 weeks? |
| No pain 0 1 2 3 4 5 6 7 8 9 10 Maximal imaginable pain |
| Seror R et al. Ann Rheum Dis doi:10.1136/annrheumdis-2013-204615 |

#### 11.3.5. Histology

### Histology

Two types of histology analysis will be conducted:

- 1. H&E
- 2. Immune Histochemistry (IHC)

Each analysis will be performed by two operators (blinded to the outcome of other's assessments). Average values will be calculated and reported.

Immune Histochemistry

(IHC)

The following parameters will be collected:

- Focus Score H&E
- Volume Fraction
- CD3/CD20 (T cell / B cell; double staining)
- CD21 (Germinal Centres)
- CD138 (plasma cells)
- IgG (B cell activity)
- IgM (B cell activity)
- IgA (B cell activity)
- Ki67 (proliferation)

Volume fraction = aggregate area / total glandular area

11.3.6. **Laboratory Biomarkers of Disease Activity** 

### **Laboratory Biomarkers of Disease Activity**

Laboratory Biomarkers of Disease Activity include (LBTESTCD):

- Serum bicarbonate (LBTESTCD=HC03\_PLC)
- Serum chloride (LBTESTCD=CL PLC)
- Cryoglobulin (LBTESTCD=CYRO\_PLG)
- Urinary Protein creatinine radio (PRTCRT\_URQ)
- Total Immunoglobulin (LBTESTCD=IG-PLC)
- IgG (LBTESTCD=IGG\_PLC)
- IgA (LBTESTCD=IGA\_PLC)
- IgM (LBTESTCD=IGM PLC)
- Serum Monoclonal Protein Electrophoresis (LBTESTCD=MPROTE\_PLC)
- Complement component 3 (LBTESTCD=C3\_PLC)
- Complement component 4 (LBTESTCD=C4\_PLC)

- Anti-Sjogrens-syndrome-related antigen A (qualitative) (LBTESTCD=SJSSAA\_PLG)
- Anti-Sjogrens-syndrome-related antigen B (qualitative) (LBTESTCD=SJSSAB\_PLG)
- Serum creatinine (LBTESTCD=CRT\_PLC)
- Urea/BUN (LBTESTCD=UREA\_PLC)
- Glomerular filtration rate (MDRD)
- Creatine kinase (LBTESTCD=CK\_PLC)
- Haemoglobin (LBTESTCD=HB\_PLC)
- White blood cell count (LBTESTCD=WBC\_PLC)
- Neutrophil count (LBTESTCD=NEUT\_BLC)
- Lymphocyte count (LBTESTCD=LYMPH\_BLC)
- Platelet count (LBTESTCD=PLT\_PLC)

In addition to this, the ratio IgG/IgA will be derived and added to the list of labtest in the Analysis and Reporting dataset. The LBTESTCD will be IGG\_IGA\_RATIO and the derivation will simply be IgG ÷ IgA. If either value is missing or lower than LLQ then this ratio will be set to missing.

### 11.3.7. Salivary Flow Rate

### **Salivary Flow Rate**

Salivary flow rate is measured at basal and stimulated state at screening/baseline and at follow-up.

Mean of baseline and follow-up visit will be calculated separately for stimulated and basal salivary flow rate. The mean will be calculated as:

 Mean Stimulated/Basal salivary flow = (Stimulated/Basal salivary flow at baseline + Stimulated/Basal salivary flow at follow-up) ÷ 2.

If value is missing at one time point (e.g. baseline), then the rate from the other time (follow-up) will be used for the mean.

The difference of the stimulate and basal salivary flow rate will be calculated for each time point:

- Screening/baseline difference = Stimulated salivary flow rate at baseline Basal salivary flow rate at baseline
- Follow-up difference = Stimulated salivary flow rate at follow-up Basal salivary flow rate at follow-up.

If one of the rate (stimulated or basal) is missing at one time point (e.g. baseline), then the rate

from the other time (follow-up) will be used to calculate the difference. If the measure of the rate is missing at both time points, then difference will be set to missing.

The mean of difference (stimulated-basal) will be derived as follows:

 Mean difference (stimulated – basal) salivary flow = (Screening/baseline difference + Follow-up difference) ÷ 2

### 11.3.8. Lacrimal Function

### **Lacrimal Function**

The lacrimal function will be assessed using Schirmer's test. The Schirmer's test is to be performed at Baseline/Screening and Visit 2. At each time point, i) the amount of wetting of strip measured in millimetre scale, in 5 minutes ii) the time taken to complete saturation of the strip.

The ratio of strip wetted to time (i/ii) will give mm of paper wetter per minute.

Strip wet per minute = (mm of paper wet/time in seconds) x 60

The time will be given in minute seconds format and will be transformed to seconds.

This value will be summarised and to correlate with imaging parameters. If one of the values (i or ii) is missing at one timepoint then the same value from the other time point will be used to calculate the ratio for a specific eye. If the measure of the rate is missing at both time points, then ratio will be set to missing.

# 11.4. Appendix 4: Premature Withdrawals & Handling of Missing Data

### 11.4.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion (i.e. as specified in the protocol) was defined as one who completed all phases of the study including the follow up.</li> <li>Withdrawn subjects may be replaced in the study at the discretion of the sponsor.</li> </ul> |
| | All available data from subjects who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified. |

### 11.4.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: <ul> <li>These data will be indicated by the use of a "blank" in subject listing displays. Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be missing data and should be displayed as such.</li> </ul> </li> </ul> |
| Outliers | Any subjects excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

## 11.4.2.1. Handling of Missing Dates

Completely missing start or end dates will remain missing, with no imputation applied.

### 11.4.2.2. Handling of Partial Dates

| Element | Reporting Detail |
|---|---|
| Concomitant | Partial dates for any concomitant medications recorded in the CRF will be |
| Medications | imputed using the following convention: |
| | <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will<br/>be used for the month</li> </ul> |
| | <ul> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day<br/>(dependent on the month and year) and 'Dec' will be used for the month.<br/>Unless this is after the end date of study; in this case the end of study date<br/>will be used.</li> </ul> |
| | <ul> <li>The recorded partial date will be displayed in listings.</li> </ul> |
| Adverse | <ul> <li>Any partial dates for adverse events will be raised to data management. If</li> </ul> |
| Events | the full date cannot be ascertained, the following assumptions will be made: |

| Element | Reporting Detail |
|---|---|
| | <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will<br/>be used for the month.</li> </ul> |
| | <ul> <li>However, if these results in a date prior to Visit 1 and the event could<br/>possibly have occurred during study from the partial information, then the<br/>Visit 1 date will be assumed to be the start date.</li> </ul> |
| | <ul> <li>The AE will then be considered to start on-study (worse case).</li> </ul> |
| | o If the partial date is a stop date, a '28/29/30/31' will be used for the day<br>(dependent on the month and year) and 'Dec' will be used for the month.<br>Unless this is after the end date of study; in this case the end of study date<br>will be used. |
| | <ul> <li>The recorded partial date will be displayed in listings.</li> </ul> |

# 11.4.2.3. Handling of Missing Data for Statistical Analysis

Missing data will remain missing with no imputation applied for the purposes of statistical analysis.

# 11.5. Appendix 5: Values of Potential Clinical Importance

# 11.5.1. Vital Signs

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------|------------------------|-------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 85 | > 160 |
| Diastolic Blood Pressure | mmHg | < 45 | > 100 |
| Heart Rate | bpm | < 40 | > 110 |

# 11.5.2. Laboratory Values

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| | | Male | | 0.54 |
| Hematocrit | Ratio of 1 | Female | | 0.54 |
| | | $\Delta$ from BL | ↓0.075 | |
| | // | Male | | 180 |
| Hemoglobin | g/L | Female | | 180 |
| | | $\Delta$ from BL | ↓25 | |
| Lymphocytes | x10 <sup>9</sup> / L | | 0.8 | |
| Neutrophil Count | x10 <sup>9</sup> / L | | 1.5 | |
| Platelet Count | x10 <sup>9</sup> / L | | 100 | 550 |
| White Blood Cell Count (WBC) | x109/ L | | 3 | 20 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Albumin | G/L | | 30 | |
| Calcium | mmol/L | | 2 | 2.75 |
| Creatinine | umol/L | | | 1.3 X ULN |
| Creatinine | umol/L | $\Delta$ from BL | | ↑ <b>44.2</b> |
| Glucose | mmol/L | | 3 | 9 |
| Potassium | mmol/L | | 3 | 5.5 |
| Sodium | mmol/L | | 130 | 150 |
| Total CO2 | mmol/L | | 18 | 32 |

# 11.6. Appendix 6: Multicentre Studies

A summary table for subject disposition will be displayed by centre, no other outputs will be produced by centre or highlighting the recruitment by site.

# 11.7. Appendix 7: Examination of Covariates, Subgroups & Other Strata

All the reporting will be separated by subject group, i.e. by healthy volunteers and pSS subjects. Subject group would be fitted as a fixed categorical variable in the ANOVA model described in Section 7.1.1.4.

# 11.8. Appendix 8: Multiple Comparisons & Multiplicity

No adjustments for multiplicity will be required.

# 11.9. Appendix 9: Model Checking and Diagnostics for Statistical Analyses

### 11.9.1. Statistical Analysis Assumptions

# Endpoint(s) 11C-MET PET/CT parameters including but not limited to SUV<sub>peak</sub>, SUV<sub>max</sub> and SUV<sub>mean</sub>. Multiparametric MRI parameters including but not limited to diffusivity (D), microvascular volume fraction (f) and K<sub>trans</sub>. Additional quantitative parameters, if deemed appropriate. Analysis of Variance (ANOVA)

- Distributional assumptions underlying the model used for analysis will be examined by
  obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted
  values (i.e. checking the normality assumption and constant variance assumption of the model
  respectively) to gain confidence that the model assumptions are reasonable.
- If there are any departures from the distributional assumptions, alternative models will be
  explored using appropriate transformed data. Mann-Whitney U test will also be used when
  untransformed data cannot be assumed to be normal.

| ` | | |
|---|---|---|
| End | point(s) | Correlation between imaging parameters with |
| | | <ul> <li>other imaging parameters</li> </ul> |
| | | <ul> <li>salivary and tear flow</li> </ul> |
| | | <ul> <li>histological scores</li> </ul> |
| | | <ul> <li>disease activity</li> </ul> |
| | | <ul> <li>lab biomarkers of disease activity</li> </ul> |
| Anal | lysis | Pearson Correlation Coefficient |

- Both variables should be normally distributed
- Linear relationship between each of the two variables
- Homoscedasticity of the data equally distributed about the regression line.
- Alternative, non-parametric method such as Spearman rank correlation will also be reported if assumptions are violated.

# 11.10. Appendix 10 – Abbreviations & Trade Marks

# 11.10.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ADC | Apparent Diffusion Coefficient |
| AE | Adverse Event |
| ANOVA | Analysis of Variance |
| Anti-SSA/B | Anti-Sjögren's-syndrome-related antigen A/B |
| A&R | Analysis and Reporting |
| CI | Confidence Interval |
| CSR | Clinical Study Report |
| CT | Computed Tomography |
| $CV_b/CV_w$ | Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| D | Pure Diffusion Coefficient |
| D* | Pseudo Diffusion Coefficient |
| DOB | Date of Birth |
| DCE | Dynamic Contrast Enhanced |
| DP | Decimal Places |
| DW | Diffusion Weighted |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Record Form |
| ESSDAI | EULAR Sjögren's Syndrome Disease Activity Index |
| ESSPRI | EULAR Sjögren's Syndrome Patient Reported Index |
| EULAR | European League Against Rheumatism |
| f | Micro vascular volume fraction |
| FDG | Fluorodeoxyglucose |
| FRP | Females of Reproductive Potential |
| FSH | Follicle Stimulating Hormone |
| HV | Healthy Volunteers |
| IA | Interim Analysis |
| ICH | International Conference on Harmonisation |
| IDSL | Integrated Data Standards Library |
| IHC | Immune Histochemistry |
| IP | Investigational Product |
| IRE | Initial Rate of Enhancement |
| IV | Intravenous |
| K <sub>trans</sub> | Exchange Rate |
| ME | Maximal Enhancement |
| MET | Methionine |
| MRI | Magnetic Resonance Imaging |
| mSv | Millisievert |
| NRS | Numeric Rating Scale |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |

| Abbreviation | Description |
|--------------|--------------------------------------------------|
| PDMP | Protocol Deviation Management Plan |
| PET | Positron Emission Tomography |
| PK | Pharmacokinetic |
| pSS | Primary Sjögren's Syndrome |
| QC | Quality Control |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| ROI | Region of Interest |
| SAC | Statistical Analysis Complete |
| SAE | Serious Adverse Event |
| SD | Standard Deviation |
| SOP | Standard Operation Procedure |
| SUV | Standardised uptake value |
| TFL | Tables, Figures & Listings |
| TIV | Total Inflammatory Volume |
| GSK | GlaxoSmithKline |

# 11.10.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies |
|---------------------------------------------------------|
| HARP |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| SAS |

# 11.11. Appendix 11: List of Data Displays

### 11.11.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|----------------------|-------------|-------------|
| Study Population | 1.1 to 1.6 | NA |
| Pharmacodynamic | 2.1 to 2.9 | 2.1 to 2.13 |
| Pharmacokinetic | 3.1 to 3.3 | 3.1 to 3.2 |
| Safety | 4.1 to 4.5 | NA |
| Biomarker | 5.1 to 5.11 | 5.1 to 5.9 |
| Section | List | ings |
| ICH Listings 1 to 21 | | 21 |
| Other Listings | 22 t | o 47 |

## 11.11.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required an example mock-up displays provided in Appendix 12: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|------------------|--------|--------|---------|
| Study Population | NA | POP_Tn | POP_Ln |
| Pharmacodynamic | EFF_Fn | EFF_Tn | EFF_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |
| Biomarker | PD_Fn | PD_Tn | PD_Ln |

### NOTES:

 Non-Standard displays are indicated in the 'IDSL / TST ID / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

### 11.11.3. Deliverable [Priority]

| Delivery [Priority] [1] | Description |
|-------------------------|-------------------------------------|
| SAC | Final Statistical Analysis Complete |

### NOTES:

1. Indicates priority (i.e. order) in which displays will be generated for the reporting effort.

# 11.11.4. Study Population Tables

| Study F | opulation Tabl | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Disposi | ition | | | | |
| 1.1. | Safety | ES1 | Summary of Subject Disposition | | SAC |
| 1.2. | Safety | NS1 | Summary of Number of Subjects by Centre ID | | SAC |
| Populat | tions Analysed | | | | |
| 1.3. | Screened | SP1 | Summary of Study Populations | | SAC |
| Demog | raphy | | | | |
| 1.4. | Safety | DM1 | Summary of Demographic Characteristics for all Enrolled Subjects | Include summary of disease duration for pSS patients. | SAC |
| 1.5. | Safety | DM1 | Summary of Demographic Characteristics for Subjects Undergone a Scan | Include summary of disease duration for pSS patients. Exclude subjects who have not completed at least one scan. | SAC |
| 1.6. | Safety | DM6 | Summary of Race and Racial Combination | | SAC |
| Concor | Concomitant Medications and Medical Conditions | | | | |
| 1.7. | Safety | CM1 | Summary of Concomitant Medications | | SAC |

# 11.11.5. Pharmacodynamic Tables

| Pharma | Pharmacodynamic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 18F-FDG | PET/CT semi- | quantitative parar | neters | | |
| 2.1. | Safety | EFF_T1 | Summary of <sup>18</sup> F-FDG PET/CT parameters | Paginate by Parameter. Subheading 'Parameter: [name]' | SAC |
| 11C-ME | FPET/CT semi- | quantitative para | meters | | |
| 2.2. | Safety | EFF_T1 | Summary of <sup>11</sup> C-MET PET/CT parameters | Paginate by Subject group and Parameters. To include ROI, side and SE with all other summary statistics. Subheading: 'Parameter: [name]' 'Subject Group: [name]' | SAC |
| 2.3. | Safety | EFF_T4 | Point Estimate and 95% CI for <sup>11</sup> C-MET PET/CT Derived Parameters of Difference in pSS vs. HV | Analysed by Parameter (SUVmean/SUVmax/SUVpeak) and ROI. When applicable for a given ROI, the analysis will be separated by the side. Summarize Means and Differences (or Ratios) with 95% CI. | SAC |

| Pharma | Pharmacodynamic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.4. | Safety | EFF_T5 | Summary of the Posterior Distribution of the Ratio and Difference of Group Means for <sup>11</sup> C-MET PET/CT Parameter by Region | Paginate by parameter and subject group. Parameters to include: SUVpeak, SUVmax and SUVmean. First two columns for ROI and side. | SAC |
| 2.5. | Safety | EFF_T6 | Posterior Probability that the Ratio and Difference of Group Means for <sup>11</sup> C-MET PET/CT Parameter Exceeds a Certain Value, by Region | Paginate by parameter and subject group. Parameters to include: SUVpeak, SUVmax and SUVmean. First two columns for ROI and side. Ratios of interest: 1, 1.5 and 2 Difference of interest: 0 Footnote: Ratio=HV/pSS Note: Values/inequality subject to change based on data | SAC |

| Pharma | harmacodynamic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Multipa | rametric MRI q | uantitative param | eters | | |
| 2.6. | Safety | EFF_T1 | Summary of Multiparametric MRI. | Paginate by Subject group and Parameters include (median and IQR) Ktrans, D, D*, f, ADC, IRE, ME, and (Mean) lipid content and gland volume as data permits. To include ROI, side (low/high/aggregated), and SE with all other summary statistics. Parameters to include: | SAC |
| 2.7. | Safety | EFF_T4 | Point estimate and 95% CI for Multiparametric MRI Derived Parameter of Difference in pSS vs. HV | Analysed by Parameter and Region of Interest. When applicable for a given ROI, the analysis will be separated by the side of the ROI. Parameters include (median and IQR) Ktrans, D, D*, f, ADC, IRE, ME, and (Mean) lipid content and gland volume as data permits. Summarize Means and Differences (or Ratios) with 95% CI. Note: P value not included as this is not a statistically powered study | SAC |

| Pharma | Pharmacodynamic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.8. | Safety | EFF_T5 | Summary of the Posterior Distribution of the Ratio and Difference of Group Means for Multiparametric MRI Parameter by Region | Paginate by parameter and subject group. Parameters to include but not limited to: Ktrans, ADC, D, and f. For each median values will be analysed. First two columns for ROI and side. | SAC |
| 2.9. | Safety | EFF_T6 | Posterior Probability that the Ratio and Difference of Group Means for Multiparametric MRI Parameter Exceeds a Certain Value, by Region | Paginate by parameter and subject group. Parameters to include but not limited to: Ktrans, ADC, D, f and volume. For each median values will be analysed. First two columns for ROI and side. Ratios of interest: 1, 1.5 and 2 Difference of interest: 0 Footnote: Ratio=HV/pSS Note: Values/inequality subject to change based on data | SAC |

Note: The above summaries will be generated if data is available.

# 11.11.6. Pharmacodynamic Figures

| Pharma | Pharmacodynamic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| <sup>18</sup> F-FD( | PET/CT semi- | -quantitative para | meters | | |
| 2.1. | Safety | EEF_F1 | Plot of Individual <sup>18</sup> F-FDG PET/CT Parameters by ROI | Paginated by Parameter and ROI. Column panel by side. Plot Subject number along X axis and parameter value along Y axis. | SAC |
| 2.2. | Safety | EFF_F2 | Mean (+/- SE) of <sup>18</sup> F-FDG PET/CT Parameters | Paginated by Parameters and ROI. Plot Sides along X axis and Mean along Y axis. Note: If transformation is required then use median +/- IQR | |
| 2.3. | Safety | EFF_F2 | Mean (+/- 95% CI) of <sup>18</sup> F-FDG PET/CT Parameters | Paginated by Parameters and ROI. Plot Side along X axis and Mean along Y axis. Note: If transformation is required then use median +/- IQR | SAC |
| 2.4. | Safety | EFF_F7 | Ratio of SUV <sub>peak</sub> (Left/Right) Assessing Asymmetry in <sup>18</sup> F-FDG PET/CT Parameter | X-axis: Subject Y-axis: Ratio of SUVpeak(left/right) Include reference line at Y=1. Footnote: Ratio of 1 (reference line) represents complete symmetry. | SAC |

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| <sup>11</sup> C-ME | PET/CT semi | -quantitative para | imeters | | |
| 2.5. | Safety | EFF_F1 | Plot of Individual <sup>11</sup> C-MET PET/CT Parameters by ROI | Paginated by Parameter and ROI. Column panel by side. Plot Subjects along X axis and parameter value along Y axis. Colour and symbol by subject group. | SAC |
| 2.6. | Safety | EFF_F3 | Mean (+/- SE) of <sup>11</sup> C-MET PET/CT Parameters. | Paginated by Parameters and ROI. Panel by sides Plot Groups (HV/pSS) along X axis and parameter value along Y axis. Note: Difference will not be presented for this plot | SAC |
| 2.7. | Safety | EFF_F3 | Point estimate and 95% CI for <sup>11</sup> C-MET PET/CT Derived Parameter of Difference in pSS vs. HV | Page by parameter and ROI. When applicable for a given ROI, the analysis will be separated by side. Plot Subject Groups along X axis and SUV along Y axis. Subheading: 'Parameter: [parameter name]' 'ROI: [ROI name]' Footnote: Difference calculated as pSS-HV. Parameters to include: SUVpeak, SUVmax and SUVmean | SAC |

| Pharma | acodynamic: Fi | gures | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.8. | Safety | EFF_F6 | Posterior Group Means and the Difference in Group Means for <sup>11</sup> C-MET PET/CT Parameter by Region | Paginate by parameter and ROI. Panel by side where appropriate. X-axis- include group (HV pSS) and diference Footnote: Difference calculated as pSS-HV. Parameters to include: SUVpeak, SUVmax and SUVmean | SAC |
| 2.9. | Safety | EFF_F7 | Ratio of SUV <sub>peak</sub> (Left/Right) Assessing Asymmetry in <sup>11</sup> C-MET PET/CT Parameter | X-axis: Subject Y-axis: Ratio of SUVpeak(left/right) Colour and symbol by subject group Include reference line at Y=1. Footnote: Ratio of 1 (reference line) represents complete symmetry. | SAC |
| Multipa | arametric MRI o | uantitative param | eters | | |
| 2.10. | Safety | EFF_F1 | Plot of Individual Multiparametric MRI Parameters by ROI | Paginated by Parameter and ROI. Column Panel by side. Plot Subject along X axis and parameter value along Y axis. Colour and symbol by subject group. | SAC |
| 2.11. | Safety | EFF_F3 | Mean (+/- SE) Plot of MRI Parameters | Paginated by Parameters and ROI. Panel by sides Plot Groups (HV/pSS) along X axis and Parameters along Y axis. | SAC |

| Pharma | Pharmacodynamic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.12. | Safety | EFF_F3 | Point estimate and 95% CI for Multiparametric MRI Derived Parameter of Difference in pSS vs. HV | Page by Regions of Interest and MRI parameter (i.e Ktrans, D, f, ADC). When applicable for a given ROI, the analysis will be separated by side (left/right/aggregated). Plot Subject Groups along X axis and parameter along Y axis. Panel by side where appropriate. Subheading: 'Parameter: [parameter name]' 'ROI: [ROI name]' Footnote: Difference calculated as pSS-HV. | SAC |
| 2.13. | Safety | EFF_F6 | Posterior Group Means and the Difference in Group Means for Multiparametric MRI Parameter by Region | Paginate by parameter and ROI. Panel by side (include left/right/aggregated) where appropriate. X-axis- include group (HV/pSS) and difference Footnote: Difference calculated as pSS-HV. Parameters to include: Ktrans, D, f, ADC. Median will be used for each parameter. | SAC |

Note: Above figures will be produced only if data is available.

### 11.11.7. Pharmacokinetic Tables

| Pharm | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Radioa | ctivity concent | rations (static <sup>18</sup> F- | FDG and <sup>11</sup> C-MET) | | |
| 3.1. | PK | PKCT1 | Summary of <sup>11</sup> C-MET Tracer Pharmacokinetic Concentration Data | Paginated by Group and type of blood (Whole and Plasma). Group to include pSS, HV and overall. Subheading: 'Subject group: [group]' 'Blood: [blood type]' | SAC |
| Radiop | harmacokineti | parameters | | | |
| 3.2. | PK | PKPT1 | Summary of Radiopharmacokinetic Parameter – Influx Rate Constant (K <sub>i</sub> ) from <sup>11</sup> C-MET PET/CT | Paginated by Group Group to include pSS, HV and overall. Subheading: 'Subject group: [Group]' | SAC |
| 3.3. | PK | EFF_T3 | Summary of correlation between PK modelling index with <sup>11</sup> C-MET PET/CT static imaging parameters | Paginated by Group Group to include pSS, HV and overall. Subheading: 'Subject group: [Group]' Change last three column titles to 'SUVpeak' 'SUVmean' and 'SUVmax' respectively. Footnote: Parotid gland side with the highest and lowest uptake values. | SAC |

# 11.11.8. Pharmacokinetic Figures

| Pharma | Pharmacokinetic : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Radioa | ctivity concent | rations (static 18F- | FDG and <sup>11</sup> C-MET) | | |
| 3.1. | PK | PKCF1P | Plot of Individual <sup>11</sup> C-MET Tracer Pharmacokinetic Concentration-Time (Linear and Semi-Log) | Paginated by Group and type of blood (Whole and Plasma). Group to include pSS, and HV. Subheading: 'Subject group: [group]' ' Blood: [blood type]' | SAC |
| Radiop | harmacokinetio | c parameters | | | |
| 3.2. | PK | EFF_F4 | Plot of Individual Radiopharmacokinetic Parameter Influx Rate Constant (K <sub>i</sub> ) versus Standardised Uptake Value of <sup>11</sup> C-MET PET/CT | Paginate by parameters SUVpeak, SUVmean and SUVmax ROI: Parotid Gland Plot Ki along X axis and SUV parameter value along Y axis. Colour by subject group. Panel by sides – side with higher parameter values and side with lower parameter values. Include Pearson's product moment correlation | SAC |

# 11.11.9. Safety Tables

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events | | | | |
| 4.1. | Safety | AE1 | Summary of All Adverse Events by System Organ Class | Paginate by subject group | SAC |
| 4.2. | Safety | AE3 | Summary of Common Adverse Events by Overall Frequency | Paginate by subject group Footnote: Common defined as 2 or more subjects | SAC |
| 4.3. | Safety | AE15 | Summary of Common Non-Serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | Paginate by subject group Footnote: Common defined as 2 or more subjects | SAC |
| Serious | and Other Sig | nificant Adverse | Events | | |
| 4.4. | Safety | AE1 | Summary of Adverse Events Leading to Withdrawal from Study by System Organ Class and Preferred Term | Paginate by subject group | SAC |
| 4.5. | Safety | AE16 | Summary of Serious Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | Paginate by subject group | SAC |

### 11.11.10. Biomarker Tables

| Biomarker: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Disease | Activity (pSS | only) | | | |
| 5.1. | Safety | EFF_T2 | Summary of Disease Activity | List score in the following order: ESSDAI ESSPRI PtGA PhGA Oral dryness Ocular dryness | SAC |
| 5.2. | Safety | EFF_T7 | Frequency of ESSDAI Component Scores | Footnote: NA: Not Applicable – Not given as an option for the category in the questionnaire. | SAC |

| Biomai | Biomarker: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 5.3. | Safety | EFF_T3 | Summary of Correlation Between Disease Activity and Imaging Parameters | Paginate by type of Disease Activity scores. Disease activity score include: ESSDAI and ESSPRI scores Pearson's and Spearman's correlation summary to be provided in the summary table. Imaging parameter from the parotid gland, and include variable for side (high or low, or aggregated). PET/CT parameter: SUVpeak MRI parameter: Median Ktrans, D, IRE, ME, f, ADC, D*; Mean lipid content and gland volume. Subheading 'Disease Activity: [name]' | SAC |
| 5.4. | Safety | EFF_T2 | Summary of Laboratory Biomarkers of Disease Activity | Including but not limited to, SS-A, SS-B, C3, C4, CH50, CRP, cryoglobulins, RF, Immunoglobulins, protein elctrophoresi. See 11.3.6 for full list. | SAC |

| Bioma | rker: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 5.5. | Safety | EFF_T3 | Summary of Correlation Between Laboratory Biomarkers of Disease Activity and Imaging Parameters | Paginate by Laboratory biomarker type. Lab biomarkers: C3, C4 levels and IgG/IgA ratio. Pearson's and Spearman's correlation summary to be provided in the summary table. Imaging parameter from the parotid gland, and include variable for side (high or low, or aggregated). PET/CT and MRI parameter: see Table 5.3 Subheading 'Laboratory Biomarker: [name]' | SAC |
| Salivar | y gland | | | | |
| 5.6. | Safety | EFF_T2 | Summary of Basal (unstimulated) and Stimulated Salivary Flow Rate (ml/min) | Replace first column with 'Salivary Flow' and add second column 'Group'. Salivary Flow column will include Basal, Stimulated and Difference. Footnote1:' Difference for each individual calculated as stimulated-basal salivary flow at that time point.' Footnote2: 'Salivary flow rate measured in millilitres per minute (ml/min).' | SAC |

| Bioma | Biomarker: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 5.7. | Safety | EFF_T3 | Summary of Correlation Between Salivary Flow Rate and Imaging Parameters. | Paginate by salivary flow type (i.e. basil, stimulated then difference) Add column for subjects group. Pearson's and Spearman's correlation summary by subject group to be provided in the summary table. Imaging parameter from the parotid gland, and include variable for side (high or low, or aggregated). PET/CT and MRI parameter: see Table 5.3 Subheading 'Salivary Flow: [name]' Footnote: 'Difference for each individual calculated as stimulated-basal salivary flow at that time point.' Footnote2: 'Footnote: 'Salivary flow rate measured in millilitres per minute (ml/min)." | SAC |
| 5.8. | Safety | EFF_T2 | Summary of Histological Scores from Salivary Gland Biopsy | First column renamed to 'Histological Scores'. Histological scores include: Maximum lymphocyte focus score Mean lymphocyte focus score Maximum Lymphoid organisation grading Mean Lymphoid organisation grading | SAC |

| Bioma | rker: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 5.9. | Safety | EFF_T3 | Summary of Correlation Between Histological Scores with Imaging Parameters. | Paginate by type Histological score. Histological scores include: Maximum lymphocyte focus score Mean lymphocyte focus score Maximum Lymphoid organisation grading Mean Lymphoid organisation grading Pearson's and Spearman's correlation summary to be provided in the summary table. Imaging parameter from the parotid gland, and include variable for side (high or low). PET/CT and MRI parameter: see Table 5.3 Subheading 'Histological Score: [name]' | SAC |
| Non-Sa | livary Gland | | | | |
| 5.10. | Safety | EFF_T2 | Summary of Strip Length Wet per Minute (mm/min) from Schirmer's Test | Include group, side of eye (most or least), Footnote: 'Ratio calculated as length (mm) paper wet divided by time taken to wet (min). The Ratio is presented as strip length wet per minute. ' | SAC |

| Biomarker: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 5.11. | Safety | EFF_T3 | Summary of Correlation Between Length Wet per Minute (mm/min) from Schirmer's Test and Imaging Parameters. | Add column for subjects group. Pearson's and Spearman's correlation summary by subject group to be provided in the summary table. Imaging parameter from the parotid gland, and include variable for side (Left or Right). PET/CT parameter: SUVpeak Subheading 'Schirmer's test: [name]' Footnote: 'Note: Ratio calculated as length (mm) paper wet divided by time taken to wet (min). The Ratio is presented as strip length wet per minute. Note: The side of the eye for the Schiremr's test is correlated with the same side of the imaging parameter.' | SAC |

# 11.11.11. Biomarker Figures

| Biomar | Biomarker: Figures | | | | | | | | |
|---|---|---|---|---|---|--|--|--|--|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] | | | | |
| Association between clinical and imaging parameters of the salivary gland | | | | | | | | | |
| 5.1. | Safety | EFF_F4 | Plot of Basal Salivary Flow Rate vs Imaging Parameters in the Parotid Gland | Paginate by parameter. Symbol by subject group where applicable Panel plot: column for the side of gland (low, high and aggregated) PET/CT parameter: SUVpeak MRI parameter: Median Ktrans, D, IRE, ME, f, ADC, D*; Mean lipid content and gland volume. Subheading 'Imaging Parameter: [imaging technique] [parameter name]' Include Pearson's product moment correlation for each group. Footnote: 'Salivary flow rate measured in millilitres per minute (ml/min).' | SAC | | | | |
| Biomar | ker: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population IDSL / TST ID / Example Shell | | Title | Programming Notes | Deliverable<br>[Priority] |
| 5.2. | Safety | EFF_F4 | Plot of Stimulated Salivary Flow Rate vs Imaging Parameters in the Parotid Gland | Paginate by parameter. Symbol by subject group where applicable Panel plot: column for the side of gland (low, high and aggregated) PET/CT and MRI parameter: see Figure 5.1 Subheading 'Imaging Parameter: [imaging technique] [parameter name]' Include Pearson's product moment correlation Footnote: 'Salivary flow rate measured in millilitres per minute (ml/min).' | SAC |
| 5.3. | Safety | EFF_F4 | Plot of Difference (Stimulated-Basal) in Salivary Flow Rate vs<br>Imaging Parameters in the Parotid Gland | Paginate by parameter. Symbol by subject group where applicable Panel plot: column for the side of gland (low, high and aggregated) PET/CT and MRI parameter: see Figure 5.1 Subheading 'Imaging Parameter: [imaging technique] [parameter name]' Include Pearson's product moment correlation | SAC |

| Biomar | ker: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | |
| 5.4. | Safety | EFF_F4 | Plot of ESSDAI score vs Imaging Parameters in the Parotid Gland | Paginate by parameter. Panel plot: column for the side of gland (low, high and aggregated) PET/CT and MRI parameter: see Figure 5.1 Subheading 'Imaging Parameter: [imaging technique] [parameter name]' Include Pearson's product moment correlation | SAC |
| 5.5. | Safety | EFF_F4 | Plot of ESSPRI score vs Imaging Parameters in the Parotid Gland | Paginate by parameter. Panel plot: column for the side of gland (low, high and aggregated) PET/CT and MRI parameter: see Figure 5.1 Subheading 'Imaging Parameter: [imaging technique] [parameter name]' Include Pearson's product moment correlation | SAC |

| Biomar | ker: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 5.6. | Safety | EFF_F4 | Plot of Laboratory Biomarker of Disease Activity vs Imaging Parameter in the Parotid Gland | Paginate by Parameter and Laboratory biomarker type. Lab biomarkers: C3, C4 levels and IgG/IgA ratio. Panel plot: column for the side of gland (low, high and aggregated) PET/CT and MRI parameter: see Figure 5.1 Subheading: 'Imaging Parameter: [imaging technique] [parameter name]' 'Laboratory Biomarker: [name]' Include Pearson's product moment correlation | SAC |
| Associa | ation between l | histological and ir | naging parameters of the salivary gland | | |
| | | EFF_F4 | Plot of Imaging Parameters vs Histological Scores from Salivary Gland Biopsy | Paginate by parameter and histological score. Panel by side of the gland: low, high, and aggregated PET/CT and MRI parameter: see Figure 5.1 Subheading: 'Imaging Parameter: [imaging technique] [parameter name]' 'Histological Score: [name]' Include Pearson's product moment correlation | SAC |

| Biomar | ker: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Associ | ation between | lacrimal gland and | I imaging parameters | | |
| 5.8. | Safety | EFF_F4 | Plot of Imaging Parameters vs Length Wet per Minute (mm/min) | Paginate by parameter. Panel plot: column for side of gland/eye (Left and Right) Symbol by subject group where applicable ROI: Lacrimal gland . PET/CT parameter: SUVpeak Subheading: 'Imaging Parameter: [imaging technique] [parameter name]' Include Pearson's product moment correlation Note: Ratio calculated as length (mm) paper wet divided by time taken to wet (min). The Ratio is presented as strip length wet per minute. Note: The side of the eye for the Schirmer's test is correlated with the same side of the imaging parameter | SAC |

| Biomar | ker: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Assoc | iation between | imaging paramete | ers | | |
| 5.9. | Safety | EFF_F5 | Plot of Imaging Parameters vs Imaging Parameters Obtained from Different Imaging Technique. | Symbol by subject group where applicable. Panel by side of the gland: low/high/aggregated Paginate by plots type with subheading of parameters being compared: FDG (SUVmean) vs CMET(SUVmean), FDG(SUVmeak) vs CMET(SUVmeak), CMET(SUVpeak) vs CMET(SUVpeak), CMET(SUVpeak) vs MRI(Mean Lipid content) FDG(SUVpeak) vs MRI(Mean Lipid Content) MRI(Mean Lipid Content) vs MRI(Median; Ktrans, IRE, ME, D, f, D* and ADC) | SAC |

## 11.11.12. ICH Listings

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Dispos | ition | | | | |
| 1. | Screened | ES7 | Listing of Reasons for Screen Failures | | SAC |
| 2. | Safety | ES2 | Listing of Reasons for Study Withdrawal | | SAC |
| Protoc | ol Deviations | | | | |
| 3. | Safety | DV2 | Listing of Important Protocol Deviations | | SAC |
| 4. | Safety | IE3 | Listing of Subjects with Inclusion/ Exclusion Criteria Deviations | | SAC |
| Popula | tions Analysed | | | | |
| 5. | Screened | SP3 | Listing of Subjects Excluded from Any Population | | SAC |
| Demog | raphy | | | | |
| 6. | Safety | DM2 | Listing of Demographic Characteristics | | SAC |
| 7. | Safety | DM9 | Listing of Race | | SAC |
| Prior a | nd Current Med | lical conditions | | | |
| 8. | Safety | MH2 | Listing of Medical Conditions | Include family history of cardiovascular disease | SAC |
| Conco | mitant Medicati | ons | | | |
| 9. | Safety | CP_CM3 | Listing of Concomitant Medications | | SAC |
| Advers | e Events | | | | |
| 10. | Safety | CP_AE8 | Listing of All Adverse Events | | SAC |
| 11. | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events | ing of Subject Numbers for Individual Adverse Events | |

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 12. | Safety | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text | | SAC |
| Serious | s and Other Sig | nificant Adverse l | Events | | |
| 13. | Safety | AE14 | Listing of Reasons for Considering as a Serious Adverse Event | | SAC |
| 14. | Safety | AE8CP | Listing of Adverse Events Leading to Withdrawal from Study | | SAC |
| Study | procedure AEs | and SAEs | | | |
| 15. | Safety | AE8CP | Listing of Adverse Events Related to Study Procedure | This includes contrast related AEs | SAC |
| Chemis | stry | | | | |
| 16. | Safety | LB5 | Listing of Clinical Chemistry Values | | SAC |
| Hemate | ology | | | | |
| 17. | Safety | LB5 | Listing of Hematology Values | | SAC |
| Urinaly | rsis | | | | |
| 18. | Safety | UR2A | Listing of Urinalysis Data | | SAC |
| All Lab | oratory | | | | |
| 19. | Safety | LB5 | Listing of All Laboratory Data for Subjects with Any Value of Potential Clinical Concern/Potential Clinical Importance | Footnote: Contains laboratory test data for continuous test results only. | SAC |
| Vital Si | gns | | | | |
| 20. | Safety | VS4 | Listing of All Vital Signs | | SAC |
| 21. | Safety | VS4 | Listing of All Vital Signs for Subjects with any Value of Potential Clinical Importance | SAC | |

# 11.11.13. Non-ICH Listings

| Non-ICI | H : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Study P | opulation | | | | • |
| 22. | Safety | EFF_L4 | Listing of Tobacco Use | | SAC |
| 23. | Safety | EFF_L5 | Sjogren's Syndrome Disease History | Sjogren's Syndrome patients only | SAC |
| Safety | | | | | |
| 24. | Safety | EFF_L6 | Listings of Antibody Test Results | Sjogren's Syndrome patients only | SAC |
| 25. | Safety | EFF_L8 | Listing of Dental Work History | | |
| 18F-FDG | PET/CT semi- | quantitative parar | meters | | |
| 26. | Safety | EFF_L1 | Listing of <sup>18</sup> F-FDG PET/CT Parameters | | SAC |
| 11C-ME | Γ PET/CT semi | i-quantitative para | meters | | |
| 27. | Safety | EFF_L1 | Listing of <sup>11</sup> C-MET PET/CT Parameters | | SAC |
| 28. | Safety | | RAW SAS Output of Statistical Analysis Results for Difference in <sup>18</sup> F-FDG PET/CT Parameter | | SAC |
| 29. | Safety | | RAW SAS Output of Bayesian Analysis Results of <sup>18</sup> F-FDG PET/CT Parameter | | SAC |
| 30. | Safety | EFF_L7 | Listing of Totality of Meal Ingested | | |
| Multipa | rametric MRI q | uantitative param | eters | | • |
| 31. | Safety | EFF_L1 | Listing of MRI Parameters | | SAC |
| 32. | Safety | | RAW SAS Output of Statistical Analysis Results for Difference in MRI Parameter | | SAC |
| 33. | Safety | | RAW SAS Output of Bayesian Analysis Results for MRI Parameter | | SAC |

| Non-IC | H : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Contra | st Agent | | | | |
| 34. | Safety | EFF_L2 | Listings of Tracer and Contrast Agent Administration Volume | | SAC |
| Radioa | ctivity concent | rations (static 18F- | FDG and <sup>11</sup> C-MET) | | |
| 35. | PK | PKCL1P | Listing of <sup>18</sup> F-FDG Tracer Pharmacokinetic Concentration Data | Paginated by Whole Blood and Plasma | SAC |
| 36. | PK | PKCL1P | Listing of <sup>11</sup> C-MET Tracer Pharmacokinetic Concentration-Time Data | Paginated by Whole Blood and Plasma | SAC |
| Radiop | harmacokineti | Parameters | | | |
| 37. | PK | PKPL1P | Listing of Influx Rate Constant(K <sub>i</sub> ) | | SAC |
| Diseas | e index (pSS pa | atients only) | | | |
| 38. | Safety | EFF_L3 | Listing of Blood Biomarkers of Disease Activity | | SAC |
| 39. | Safety | EFF_L3 | Listing of ESSDAI Scores and Components | Include components scores then final scores – this will be a new column after 'actual time' column consisting of component names and final score. Domain score should include both the category and score (i.e. Low=2) | SAC |
| 40. | Safety | EFF_L3 | Include components scores then final | | SAC |
| 41. | Safety | EFF_L3 | Listing of Patients' Global Assessment | | SAC |
| 42. | Safety | EFF_L3 | Listing of Physician's Global Assessment (VAS 0-100mm) | | SAC |
| 43. | Safety | EFF_L3 | Listing of Oral Dryness Numeric Rating | isting of Oral Dryness Numeric Rating | |
| 44. | Safety | EFF_L3 | Listing of Ocular Dryness Numeric Rating | | |

| Non-ICI | Non-ICH : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Salivary | Gland Specifi | c Endpoints | | | |
| 45. | Safety | EFF_L3 | Listing of Basal Salivary Flow Rate (ml/min) | | SAC |
| 46. | Safety | EFF_L3 | Listing of Stimulated Salivary Flow Rate (ml/min) | | SAC |
| 47. | Safety | EFF_L3 | Listing of Histological Score from Salivary Gland Biopsy | Include a column for cell type. | SAC |
| Non-sal | Non-salivary gland | | | | |
| 48. | Safety | EFF_L3 | Listing of Paper Wetted and Time to Wet from Schirmer's Test | Include column (last) for change from baseline. | SAC |

203818

### 11.12. Appendix 12: Example Mock Shells for Data Displays

Example : EFF\_T1 Protocol : 203818


Population : Safety

Table 2.1 Summary of <sup>18</sup>F-FDG PET/CT parameters

Parameter: Parameter 1

| Region of Interest | Sides | Group | Ν | n | Mean | SD | SE | Q1 | Median | Q3 | Min. | Max. |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ROI 1 | Low | pSS<br>HV | xx<br>xx | xx<br>xx | XX.X<br>XX.X | XX.XX<br>XX.XX | XX.XX<br>XX.XX | XX.X<br>XX.X | XX.X<br>XX.X | XX.X<br>XX.X | xx<br>xx | xx<br>xx |
| | High | pSS<br>HV | xx<br>xx | xx<br>xx | XX.X<br>XX.X | XX.XX<br>XX.XX | XX.XX<br>XX.XX | XX.X<br>XX.X | XX.X<br>XX.X | XX.X<br>XX.X | xx<br>xx | xx<br>xx |
| ROI 2 | NA | pSS | Xx<br>xx | Xx<br>xx | XX.X<br>XX.X | XX.XX<br>XX.X | XX.XX | XX.X | XX.X | xx.x | xx | Xx |

Note: NA: Sides are not applicable for all ROI.

Programming Note: Include Groups as a separate column next to Sides for 11C-MET PET/CT parameters summary.

Example : EFF\_T2 Page 1 of n

Protocol : 203818 Population : Safety

Table X.X

Summary of Disease Activity (pSS only)

Disease Activity N n Mean SD Median Minimum Maximum

ESSDAI score

ESSRPI score

Patient Global assessment (VAS)

Physician Global Assessment (VAS)

Oral dryness numerical rating

Ocular dryness numerical rating

: EFF\_T3 : 203818 Page 1 of n Example

Protocol Population : Safety

Table x.x

Summary of Correlation Between Disease Activity and Imaging Parameters

Disease Activity: [name of index]

| Scan / Parameter | Side | Pearson's correlation / 95% CI | Spearman's correlation / 95% CI |
|---|---|---|---|
| TIC-MET / | High | x.xx / | x.xx / |
| SUVpeak | Low | (x.xx, x.xx)<br>x.xx / | (x.xx, x.xx)<br>x.xx / |
| F-FDG /<br>SUVpeak | High<br>Low | (x.xx, x.xx)<br>x.xx /<br>(x.xx, x.xx)<br>x.xx /<br>(x.xx, x.xx) | (x.xx, x.xx)<br>x.xx /<br>(x.xx, x.xx)<br>x.xx /<br>(x.xx, x.xx) |
| MRI /<br>Ktrans | High<br>Low | x.xx /<br>(x.xx, x.xx)<br>x.xx /<br>(x.xx, x.xx) | x.xx /<br>(x.xx, x.xx)<br>x.xx /<br>(x.xx, x.xx) |

Example: EFF\_T4
Protocol: 203818
Population: Safety

Protocol: 203818 Page 1 of n

Table x.xx

Point estimate and 95% CI for [imaging method] Derived Parameter of Difference in pSS vs. HV 95% CI for

| ROI: [ | | ] | Side: [ | ] | | | - 1 0 0 | -1.05 |
|---|---|---|---|---|---|---|---|---|
| N | Group | | | n | Mean | Standard<br>Error | Difference<br>from HV | Difference<br>(Lower, Upper) |
| XX | HV | | | XX | x.xx | x.xxx | | |
| XX | pSS | | | XX | X.XX | X.XXX | X.XX | (x.xx, x.xx) |
| XX | HV | | | XX | x.xx | x.xxx | | |
| XX | pSS | | | XX | X.XX | X.XXX | X.XX | (x.xx, x.xx) |

Example: EFF\_T5
Protocol: 203818
Population: Safety


### Summary of the Posterior Distribution of the Ratio and Difference of Group Means for [Imaging method] parameters by Region

| | | | | | | | Posterior d | istribution _ | | <del></del> |
|---|---|---|---|---|---|---|---|---|---|---|
| Parameter | ROI | Group | Prior Distribution for<br>Θ | Value of σ<br>used in then<br>model | Mean | SD | Median | 25th<br>quartile | 75th<br>quartile | 95% Credible Interval |
| Mean SUV | Parotid Gland | pSS (N=xx) | normal(0, sd = 100) | 1 | x.xx | x.xx | x.xx | X.XX | X.XX | (x.xx,x.xx) |
| | | HV (N=xx) | normal(0, sd = 100) | 1 | x.xx | x.xx | x.xx | x.xx | x.xx | (x.xx,x.xx) |
| | | Difference | | | | | | | | |
| | | | | | x.xx | x.xx | x.xx | x.xx | x.xx | (x.xx,x.xx) |
| | | Ratio | | | | | | | | |
| | | | | | x.xx | x.xx | x.xx | x.xx | x.xx | (x.xx,x.xx) |
| | Submandibular<br>Gland | | | | | | | | | |

pSS=primary Sjogren's Syndrome patients HV=Health Volunteers, ROI = Region of Interest


203818

Number of MCMC iterations, excluding the burn-in iterations = 5,000. Number of burn-in iterations = 10,000 The PET parameters are assumed to follow a normal distribution with unknown mean  $\Theta$  and known variance  $\sigma^2$  (i.e.  $N(\Theta, \sigma^2)$ ). Difference calculated as pSS-HV and ratio as pSS/HV. 95% credible intervals based on the highest posterior density interval.

Example: EFF\_T6
Protocol: 203818
Population: Safety


Posterior Probability that the Ratio and Difference of Group Means for [Imaging Method] Parameter Exceeds a Certain Value, by Region

| Parameter (units) | Region | P(ratio) > 0.5 | P (ratio) > 1 | P(ratio) > 1.5 | P(Difference) > 0 |
|---|---|---|---|---|---|
| Mean SUV | | | | | |

Note: P(ratio) > 1 is the probability that the posterior ratio of group means exceeds 1 based on 5,000 simulated posterior predicted values. Ratio of pSS patients to Healthy Volunteers and difference of pSS-HV.

Example : EFF\_T7
Protocol : 203818
Population : Safety


 $\label{eq:continuous} \begin{tabular}{ll} Table X.X \\ \begin{tabular}{ll} Summary of ESSDAI Component Scores \\ Activity Level \\ \end{tabular}$ 

| Domain | No | Low | Moderate | High |
|-----------------|------|------|----------|------|
| Constitutional | n(%) | n(%) | n(%) | NA |
| Lymphadenopathy | n(%) | n(%) | n(%) | n(%) |
| Glandular | n(%) | n(%) | n(%) | NA |
| Articular | n(%) | n(%) | n(%) | n(%) |
| Cutaneous | n(%) | n(%) | n(%) | n(%) |
| Pulmonary | n(%) | n(%) | n(%) | n(%) |


| n(%) | n(%) | n(%) | n(%) |
|---|---|---|---|
| n(%) | n(%) | n(%) | n(%) |
| n(%) | n(%) | n(%) | n(%) |
| n(%) | NA | n(%) | n(%) |
| n(%) | n(%) | n(%) | n(%) |
| n(%) | n(%) | n(%) | NA |
| | n(%) n(%) n(%) n(%) | n(%) n(%) n(%) n(%) n(%) NA n(%) n(%) | n(%) n(%) n(%) n(%) n(%) n(%) n(%) NA n(%) n(%) n(%) n(%) |

Example : EFF\_L1 Protocol : 203818

: Safety

Population


Listing xx Listing of <sup>18</sup>F-FDG PET/CT Parameters

**Imaging Parameter** 

| Subject | ROI | SUV mean | SUV peak | $SUV_{\text{max}}$ | TR | TIV |
|---|---|---|---|---|---|---|
| xxxxx | Parotid Left | | | | | |
| | Parotid<br>Right | | | | | |

**SUV**= Standardised Uptake Value, TR = tissue-to-reference ratio ,TIV = total inflammatory volume.(description of all Parameter)

\_

.

Example Protocol

Population

: EFF\_L2 : 203818 : Safety


Listing No. XX

Listing of Tracer and Contrast Agent Administration Volume

| Subjid | Visit | Contrast<br>Agent/Tracer | Volume of Administration (Unit) |
|--------|--------|--------------------------|---------------------------------|
| XXX | Visit1 | Gadolinium | X |
| | Visit1 | C-MET | X |
| | Visit2 | FDG | X |

Example: EFF\_L3
Protocol: 203818
Population: Safety


Listing X
Listing of Patients' Global Assessment (VAS 0-100mm)

| Subj | Planned<br>Relative<br>Time | Actual | date <mark>/time</mark> | Study<br>Day | Score |
|---|---|---|---|---|---|
| PPD | Baseline | PPD | /14:00:00 | 1 | 100 |
| | Baseline | | /14:00:00 | 1 | 98 |

EFF\_L4 203818

Listing 22 Listing of Tobacco Use

Example:
Protocol:
Population:

| Site ID/<br>Subject ID | Smoking history | Last smoke | Average cigarettes per day | Safety |
|---|---|---|---|---|
| XX/XXXXX | Never | NA | | |
| XX/XXXXX | Current | NA | | |
| XX/XXXXX | Former | YYYY-MM-DD | | |

Example: EFF\_L5
Protocol: 203818

Population:

Listing 23
Sjogren's Syndrome Disease History


| Site ID/<br>Subject ID | Date of Formal pSS Diagnosis | Duration since<br>Formal Diagnosis<br>(months) | Classification |
|---|---|---|---|
| XX/XXXXX | YYYY-MM-DD | XX.X | Ocular symptoms Oral symptoms |
| XX/XXXXX | YYYY-MM-DD | xx.x | Histopathology<br>Salivary gland<br>involvement |
| XX/XXXXX | | | |

Example: EFF\_L6
Protocol: 203818

Population:

Listing 24 Listing of Antibody Test Result


| Site ID/ | Date of | | |
|------------|------------|----------|-----------|
| Subject ID | assessment | Test | Result |
| XX/XXXXX | YYYY-MM-DD | Total Ig | X.XX |
| | | IgG | X.XX |
| | | IgA | X.XX |
| | | IgM | No result |
| XX/XXXXX | YYYY-MM-DD | Total Ig | X.XX |
| | | IgG | X.XX |
| | | IgA | X.XX |
| | | IgM | No result |
| XX/XXXXX | | | |

Example: EFF\_L7
Protocol: 203818

Population:

#### Listing 28 Listing of Totality of Meal Ingested


| Site ID/<br>Subject ID | Meal start time | Meal end time | Duration | Meal<br>ingested |
|---|---|---|---|---|
| XX/XXXXX | HH:MM | нн:мм | x.xx | 1-25% |
| xx/xxxxx | HH:MM | HH:MM | x.xx | 76-100% |
| XX/XXXXX | нн:ММ | HН:MM | x.xx | Yes |

| Example: | EFF_L8 | |
|----------|--------|---|
| _ | | _ |

Protocol:  $20\overline{3}818$ 

Population:

| Site ID/<br>Subject ID | Dental Work | Yes/No - Location_ | Page 1 of n |
|---|---|---|---|
| XX/XXXXX Non-metallic filling or crowns | | No | Safety |
| | Other fillings | Yes - Top Left | |


Example : EFF\_F1
Protocol : 203818
Population : Safety

Figure 2.2 Plot of Peak Standardised Uptake Value (SUV $_{\rm peak}$ ) from  $^{18}{\rm F-FDG}$  PET/CT by ROI

ROI: Parotid Gland





Programming Note: Panel plot when the ROI is split by side (above) otherwise single plot (below)




Example : EFF\_F2
Protocol : 203818
Population : Safety

Figure 2.x Mean (+/- SE) of <sup>18</sup>F-FDG PET/CT Parameters.

Parameter: [Parameter 1] ROI: [ROI 1]



Example : EFF\_F3 Page 1 of 1

Protocol : 203818 Population : Safety

Figure 2.x

Point estimate and 95% CI for [imaging method] derived parameters of Difference in pSS vs. HV Parameter: [Parameter 1] ROI: [ROI 1]

Side: Low Side: High





Example : EFF\_F4 Page 1 of n

Protocol : 203818
Population : Safety

Figure x.x

Plot of Disease Activity scores vs Imaging Parameters in the Parotid Gland

Parameter: SUVpeak Disease Activity: ESSDAI score



r: Pearson's product moment correlation



Example : EFF\_F5 Protocol : 203818 Page 1 of n

Protocol : 203818 Population : Safety

Plot of Imaging from Different Imaging

Figure x.x

Parameters vs Imaging Parameters Obtained Technique.

Parameter: C-MET(SUVpeak) vs F-FDG (SUVpeak)



r: Pearson's product moment correlation

Example : EFF\_F6 Page 1 of n

Protocol : 203818
Population : Safety

Figure x.x
Posterior Group Means and the Difference in Group Means for [Imaging method] Parameter by Region



Example : EFF\_F7
Protocol : 203818
Population : Safety

Figure x.x
Ratio of SUV<sub>peak</sub> (Left/Right) Assessing Asymmetry in <sup>11</sup>C-MET PET/CT Parameter



Ratio of 1 (reference line) represents complete symmetry.